

# Statistical Analysis Plan (SAP) to the JC-02 Protocol August 8, 2019

A Prospective, Multicenter, Randomized, Study of the Safety and Efficacy of Intravitreal Injection of Human Retinal Progenitor Cells (jCell) in Adult Subjects with Retinitis Pigmentosa (RP)

NCT03073733



## Statistical Analysis Plan

## jCyte, Inc. Protocol JC-02

## A Prospective, Multicenter, Randomized, Study of the Safety and Efficacy of Intravitreal Injection of Human Retinal Progenitor Cells (jCell) in Adult Subjects with Retinitis Pigmentosa (RP)

Protocol Version: Amendment 7 (March 19, 2018)

**Sponsor:** jCyte, Inc

2549 East bluff Drive, Suite 196 Newport Beach, CA 92660

Prepared by:

Synteract 430 Davis Drive Morrisville, NC 27560

| Version | Date |
|------------|------------|
| V0.1 | 18Apr2019 |
| V0.2 | 04Jun2019 |
| V0.3 | 19Jun2019 |
| V0.4 | 03Jul2019 |
| V1.0 Final | 16July2019 |
| V2.0 Final | 08Aug2019 |

# Approval

Upon review of this document, including table, listing, and figure shells, the undersigned approves the Statistical Analysis Plan. The analysis methods and data presentation are acceptable.

| Signature | Date |
|----------------------------------|----------|
| | <u> </u> |
| • | |
| S Y n teract | |
| BRINGING CLINICAL TRIALS TO LIFE | |

## TABLE OF CONTENTS

| LIS | T OF | ABBREVIATIONS | 5 |
|-----|-------|--------------------------------------------------------|----|
| DE | FINIT | TIONS | 7 |
| 1. | INTF | RODUCTION | 8 |
| | 1.1 C | HANGES FROM PROTOCOL | 8 |
| 2. | STUI | DY OBJECTIVES | 8 |
| | | RIMARY OBJECTIVE | |
| | | ECONDARY OBJECTIVE | |
| 3. | | DY DESIGN AND PLAN | |
| 4. | | ERMINATION OF SAMPLE SIZE | |
| 5. | GEN | ERAL ANALYSIS CONSIDERATIONS | 10 |
| 6. | ANA | LYSIS POPULATIONS | 10 |
| 7. | STUI | DY POPULATION | 11 |
| | 7.1 | SUBJECT DISPOSITION | |
| | 7.2 | PROTOCOL DEVIATIONS | |
| | 7.3 | DEMOGRAPHIC AND BASELINE CHARACTERISTICS | 12 |
| | 7.4 | PRIOR AND CONCOMITANT MEDICATIONS | 12 |
| 8. | EFFI | ICACY ANALYSES | 12 |
| | 8.1 | EFFICACY VARIABLES | 12 |
| | 8.2 | BASELINE VALUES | 13 |
| | 8.3 | HANDLING OF DROPOUTS OR MISSING DATA | |
| | 8.4 | INTERIM ANALYSIS AND DATA MONITORING | |
| | 8.5 | EXAMINATION OF SUBGROUPS | |
| | 8.6 | MULTIPLE COMPARISON/MULTIPLICITY | |
| | 8.7 | MULTICENTER STUDIES | |
| 9. | MET | THODS OF EFFICACY ANALYSIS | |
| | 9.1 | BEST CORRECTED VISUAL ACUITY (BCVA) | |
| | 9.2 | VISUAL FIELD EXAMINATION | |
| | 9.3 | MOBILITY | |
| | 9.4 | CONTRAST SENSITIVITY (CS) | |
| | 9.5 | Low Vision Visual Functional Questionnaire (LV-VFQ 48) | |
| 10. | SAFI | ETY ANALYSES | |
| | 10.1 | STUDY DRUG ADMINISTRATION | |
| | 10.2 | ADVERSE EVENTS | |
| | 10.3 | CLINICAL LABORATORY EVALUATION | |
| | | VITAL SIGNS | |
| | | PHYSICAL EXAMINATION | |
| | 10.6 | OPHTHALMIC AES | 23 |

| | 10.6.1 SLIT LAMP AND FUNDUS PHOTOGRAPHY | 23 |
|-----|-----------------------------------------------------------------|----|
| | 10.6.2 Intraocular Pressure (IOP) | 23 |
| | 10.6.3 B-SCAN | |
| | 10.6.4 DILATED FUNDOSCOPIC EXAMINATION | 23 |
| | 10.6.5 Post Injection Clinical Vitreous Exam | 24 |
| | 10.6.6 OPTICAL COHERENCE TOMOGRAPHY (OCT) | 24 |
| | 10.7.7 AUTOFLUORESCENCE | 24 |
| 11. | REFERENCES | 24 |
| | APPENDIX A: PRESENTATION OF DATA AND PROGRAMMING SPECIFICATIONS | 25 |
| | APPENDIX B: LIST OF TABLES, FIGURES, AND LISTINGS | 28 |
| | APPENDIX C: TABLE LAYOUTS | |
| | APPENDIX D: LISTING LAYOUTS | 72 |

## LIST OF ABBREVIATIONS

AE Adverse Event

ATC Anatomical Therapeutic Chemical

BCVA Best Corrected Visual Acuity

BP Blood Pressure bpm Beats per Minute

CIL Critical Illumination Level

cm Centimeter(s)
CRF Case Report Form
CS Clinically Significant
CS Contrast Sensitivity
CSR Clinical Study Report

CTCAE Common Terminology Criteria for Adverse Events

DDT Dictionary Derived Term
DRA Donor Reactive Antibody

EE Efficacy Evaluable

E-ETDRS Electronic Early Treatment for Diabetic Retinopathy Study

ERG Electroretinogram EZ Ellipsoid Zone

FrACT Freiburg Visual Acuity & Contrast Test

FST Full Field Scopic Threshold hRPC Human Retinal Progenitor Cells

ICH International Conference on Harmonization

in Inch(es)

ITT Intent-to-Treat kg kilogram(s)

LOD Limit of Detection

LogMAR Logarithm of minimal angle of resolution LV-VFQ48 Low Vision Functional Questionnaire

mITT Modified Intent-to-Treat

msec Millisecond

MSS Maximum Step Speed

MedDRA Medical Dictionary for Regulatory Activities

mg Milligram(s)

mmHg Millimeter of Mercury NCS Not Clinically Significant

OCT Optical Coherence Tomography

OD Oculus Dextrus (right eye)
OS Oculus Sinister (left eye)
PRA Panel Reactive Antibody

PT Preferred Term

RP Retinitis Pigmentosa
SAE Serious Adverse Event
SAP Statistical Analysis Plan

SD Standard Deviation SOC System Organ Class

TEAE Treatment-Emergent Adverse Event

TLs Tables and Listings

VFQ-48 Visual Function Questionnaire WHO World Health Organization

## **DEFINITIONS**

Adverse Event An adverse event (AE) is any reaction, side effect, or

other untoward event, regardless of relationship to study

drug, which occurs anytime during the study.

Intent-to-Treat Population

(ITT)

All randomized subjects who provide any post-

randomization data.

Modified Intent-to-Treat Population (mITT)

All randomized subjects who provide any postrandomization data, excluding subjects with missing baseline values or who are unable to perform the relevant assessment at baseline. mITT populations will be defined

for each secondary endpoint using this criteria.

Efficacy Evaluable Population (EE)

All randomized subjects who provide any postrandomization data, excluding subjects with missing baseline values. The LOD will be used as the baseline value for subjects who are unable to perform the relevant assessment at baseline. Subjects for whom baseline is completely missing will be considered nonevaluable for the relevant endpoint.

Safety Population

All subjects who received any amount of study drug.

Serious AE

An AE occurring at any dose that: results in death; is a life-threatening experience; requires inpatient hospitalization or prolongation of an existing hospitalization; results in a persistent or significant disability/incapacity; or is a congenital anomaly/birth defect in the offspring of a subject who received study

drug.

Treatment-emergent AE

AEs that occur after the study treatment (injection or

sham injection)

#### 1. INTRODUCTION

This document outlines the statistical methods to be implemented during the analyses of data collected within the scope of jCyte Protocol JC-02 [A Prospective, Multicenter, and Randomized, study of Safety and Efficacy of Intravitreal injection of Human Retinal Progenitor Cells (jCell) in Adult Subjects with Retinitis Pigmentosa (RP)]. The purpose of this plan is to provide specific guidelines from which the statistical analyses will proceed. Any deviations from this plan will be documented in the clinical study report (CSR).

## 1.1 Changes from Protocol

Per the protocol section 10.2.2, subjects who cannot perform a specific visual test at baseline (e.g. mobility) will be considered nonevaluable for analysis of that assessment. In this SAP, patients who can't perform a visual test are included using the value determined to be the Limit of Detection (LOD).

#### 2. STUDY OBJECTIVES

## 2.1 Primary Objective

The primary objective is to assess the changes in visual function as measured by BCVA at 12 months following a single injection of jCell at one of two dose levels (Test) compared to sham-treated controls in a cohort of adult subjects with RP with baseline best corrected visual acuity (BCVA) in the study eye equal to or worse than 20/80 and no worse than 20/800.

## 2.2 Secondary Objective

The secondary objectives of the study are

- To assess the impact of jCell injection at two dose levels based on visual function (VF, CS) and functional vision (mobility, VA LV VFQ-48).
- To evaluate the safety and tolerability of jCell injection in subjects with RP.

## 3. STUDY DESIGN AND PLAN

This is a prospective, multicenter, randomized, single-masked, three-arm, Phase 2b trial of human retinal progenitor cells (jcell) for the treatment of retinitis pigmentosa (RP). Study subjects will be screened for eligibility and informed consent will be obtained

## Randomization and Masking:

Up to 85 subjects will be randomized 1:1:1 to one of two Test (jCell treatment) arms (3 x 10<sup>6</sup> jCell dose or 6 x 10<sup>6</sup> jCell dose) or to the Control (sham-treated) study group. Study subjects will be masked with respect to which treatment they are receiving, although study investigators and those involved in certain aspects of treatment and assessment (where injected cells are visualized) cannot feasibly be masked. However, site staff that perform key assessments (primary and secondary efficacy endpoints) will be masked to the treatment assignment. Assessors will be told which eye is the study eye for each subject but will not know whether that subject is assigned to a Test or Control group. Once the subject has completed 12 months of follow up, that subject may request to have his/her treatment revealed. If the subject was assigned to the control group, the subject will be offered the opportunity to cross over to the test group, and will be randomized to one of the two dose levels. Although all cross over subjects will receive Test treatment, the same masking procedures will be in place during the crossover portion so as to mask the dose level to which the subject was assigned.

## **Study Population:**

The phase 2b study design is focused on subjects with visual acuity of 20/80 or worse in the study eye, without macular edema, and whose quality of life is already negatively impacted by the disease to a large degree. The cut-off of 20/80 for the study eye was selected to provide a sufficient "margin" for observation of potential benefit, as measured in terms of gains in BCVA.

Subjects randomized to one of the Test groups will receive a single intravitreal injection of either 3 x  $10^6$  jCell dose or 6 x  $10^6$  jCell into the study eye. Subjects randomized to Control group will not receive treatment, but will undergo a similar procedure that is a sham injection in the study eye. Subjects in both cohorts will be followed for one year for safety and evidence of jCell effects.

## 4. DETERMINATION OF SAMPLE SIZE

The sample size of 25 subjects per treatment arm is needed to achieve the targeted level of statistical power; the trial could enroll up to 85 subjects if needed to address irregularities in trial conduct or potential drop-outs. Assume the standard deviation for the 12-month change in BCVA is 5 letters. Then, for each pairwise comparison with the control group, a randomized trial with 25 patients per arm will have 90% power to detect a true treatment effect of a mean of 5 letters, when using a t-test having (one-sided) 0.0125 false positive error rate.

## 5. GENERAL ANALYSIS CONSIDERATIONS

The statistical analyses will be reported using summary tables and listings (TLs). The International Conference on Harmonization (ICH E3) numbering convention will be used for all TLs. unless otherwise noted, all statistical testing will be 2-sided and will be performed at the 0.05 significance level. Tests will be declared statistically significant if the calculated P value is  $\leq 0.05$ . Continuous variables will be summarized with means, standard deviations, medians, minimums, and maximums. Categorical variables will be summarized by counts and by percentage of subjects in corresponding categories. Percentages for missing values are omitted and do not account for the percent calculation of other categories. Percentages are routinely based on the total category count excluding the missing category if not otherwise mentioned. Percentages showing a rate relative to the total number of subjects in this group are given in special tables (e.g. AE tables). Footnotes will specify the percent basis. All summary tables will be presented by dose level (3 x  $10^6$  jCell dose, 6 x  $10^6$  jCell and sham). Unless otherwise noted, the baseline value will be the last non-missing value recorded prior to the first dose of study drug.

Individual subject data obtained from the case report forms (CRFs) and derived data will be presented by subject in data listings.

The analyses described in this plan are considered *a priori*, in that they have been defined prior to database lock. Post-hoc analyses will be labeled as such on the output and identified in the CSR.

All analyses and tabulations will be performed using SAS® Version 9.4 or higher. Tables, listings, and figures will be presented in RTF format. Upon completion, all SAS® programs will be validated by an independent programmer. In addition, all program output will undergo a senior level statistical review. The validation process will be used to confirm that statistically valid methods have been implemented and that all data manipulations and calculations are accurate. Checks will be made to ensure accuracy, consistency with this plan, consistency within tables, and consistency between tables and corresponding data listings. Upon completion of validation and quality review procedures, all documentation will be collected and filed by the project statistician or designee.

#### 6. ANALYSIS POPULATIONS

The following subject population will be used for safety analyses:

Safety population will include all subjects who receive any study treatment (including sham).

The following subject population will be used for efficacy analyses:

- Intent-to-Treat (ITT) population will include all subjects enrolled and randomized in the study and who provide any post-randomization data. Subjects for whom randomization assignment is noted in the clinical database will be considered to be enrolled in the study.
- Modified Intent-to-Treat (MITT) population will be defined as all randomized subjects who provide any post-randomization data, excluding subjects with missing baseline or who are below the LOD at baseline. mITT populations will be defined for each secondary endpoint using this criteria
- An Efficacy Evaluable (EE) population will be defined for each secondary
  endpoint where all randomized subjects who provide any post-randomization
  data, including subjects who are below the LOD at baseline (e.g. unable to
  perform the assessment). The LOD will be used as the baseline value for subjects
  unable to perform the assessment. Subjects for whom baseline is completely
  missing will be considered nonevaluable for the relevant endpoint...

## 7. STUDY POPULATION

## 7.1 Subject Disposition

Subject disposition information will be summarized for all subjects by dose level (3 x  $10^6$  jCell dose, 6 x  $10^6$  jCell dose and Sham). Summaries will include: the number of enrolled subjects, the number of subjects in each analysis population, and the primary reason for discontinuation.

#### 7.2 Protocol Deviations

Major protocol deviations that could potentially affect the efficacy or safety conclusions of the study will be identified prior to database lock. Major protocol deviations may include, but are not limited to:

- Subjects who did not satisfy selected inclusion and exclusion criteria;
- Subjects who received the incorrect dose;
- Subjects who received an excluded concomitant treatment.

All protocol deviations will be presented in a listing by dose level and deviation category,

## 7.3 Demographic and Baseline Characteristics

Demographic variables include: age, sex, ethnicity and race. Age will be calculated in years relative to the informed consent date. Other baseline characteristics include: medical history, ocular medical history, height, weight, and study eye (OD [right] or OS [left]).

Descriptive statistics will be presented for age, height, and weight. Frequency counts and percentages will be presented for sex, ethnicity, race, study eye, ocular medical history. Demographic and baseline characteristics will be summarized for the Safety and ITT populations. If Safety and ITT populations are identical, the two tables will be combined into a single summary.

Ocular medical history (OMH) or Medical history condition or event will be mapped to primary System Organ Class and dictionary-derived term by using MedDRA 20.0.

Medical history and Ocular medical history will be presented in a listing.

#### 7.4 Prior and Concomitant Medications

Prior and concomitant medication verbatim terms on case report forms (CRFs) will be mapped to Anatomical/Therapeutic/Chemical (ATC) class and Preferred Names using the World Health Organization (WHO) Drug Dictionary Enhanced (version March 1, 2017)...

Prior and concomitant medications will be presented in a listing.

## 8. EFFICACY ANALYSES

The primary efficacy analysis will be based on the ITT population.

#### 8.1 Efficacy Variables

The response to jCell injection will be assessed based on the following:

Best Corrected Visual Acuity (BCVA): BCVA will be measured with the
electronic visual acuity testing algorithm (E-ETDRS). For each time point
assessed, the total number of letters correct using E-ETDRS will be recorded for
each eye and recorded on the Best Corrected Visual Acuity (BCVA) case report
form. For eyes with vision worse than the upper limits of the E-ETDRS, the

Freiburg Visual Acuity & Contrast Test (FrACT) system will be used and the resultant Snellen acuity will be recorded and later converted to relevant data (e.g, letters correct.).

- Kinetic Visual Field Total Area: information regarding area in degrees squared of individual isopters or islands of vision in each eye will be recorded. Instrument target size will also be recorded as three sizes were used (V4e, III4e, and I4e) in individuals with near normal V4e isopters. In addition, observed fixation stability on a scale of 1 to 5 is recorded related to subject ability to hold fixation on a target during the entirety of kinetic field testing. Comments regarding corrective lenses used, difficulty of testing (related to reliability) and description of areas of seeing or non-seeing that are too small for mapping will be included.
- Mobility: Testing is conducted monocular (one eye at a time). Information
  regarding whether a subject is Dark Adapted, Dark Adapt start time and end time,
  Maximum step speed, Critical illumination level, and comments will be recorded
  on CRF.
- Contrast Sensitivity (CS): For each eye, Thresholds CS values will be recorded for spatial frequencies from the following range: 0.25, 0.5, 1.0, 2.0, 4.0, 8.0 and 12.0 (not all frequencies will be tested for each eye; frequency of 12 was not used).
- Low Vision Visual Functional Questionnaire (LV VA VFQ-48): Scale scores for Visual Ability, Reading, Mobility, Visual Information, and Visual Motor will be recorded on CRF. Time to complete the questionnaire and comments regarding the testing process will be recorded.

#### 8.2 Baseline Values

For efficacy variables, baseline is defined as the value obtained at baseline visit or if subject is unable to perform a secondary endpoint, a value that is determined to be the limit of detection will be used. For BCVA, if the value is missing on baseline visit, the baseline value will be the value at the screening visit.

## 8.3 Handling of Dropouts or Missing Data

For certain variables that are measured by instrument, some values are not captured exactly as the true value falling below the detection limit of the instrument. Observations that are lost due to LOD represent partial information, i.e. the value is known to be below

a certain value but otherwise unknown. The LOD values will be used for these observations unless otherwise specified. For data that is not obtained at all due to lack of assessment or missed visits it is assumed that the data is close to missing at random after accounting for terms in the model. The key analysis for all variables will exclude the truly missing variable and will involve no imputation. Sensitivity analyses will involve some form of multiple imputation. No imputation is consistent with data that is missing at random. Multiple imputation uses the structure of the observed data along with a random component to generate multiple plausible datasets, which are analyzed individually, summarized, and then combined to produce a final result.

## 8.4 Interim Analysis and Data Monitoring

There is no planned interim analysis for the JC-02 study, however it should be noted that the study will be ongoing (cross over phase) at the time of the primary analysis, as defined in the protocol. This SAP does not include analysis involving cross over portion of the study, which will be included in an amendment. Thus the analysis of the cross over period data will be provided as an addendum to the study report.

## 8.5 Examination of Subgroups

There are no planned subgroup analyses for this study.

## 8.6 Multiple Comparison/Multiplicity

No adjustments for multiplicity will be made in this study.

#### 8.7 Multicenter Studies

Analyses to compare differences in response by center or any treatment by center interactions are not planned.

#### 9. METHODS OF EFFICACY ANALYSIS

Descriptive statistics will be used to tabulate and summarize study outcomes. Results of clinical testing of the non-injected eye will also be described. Changes from baseline in the treated groups will be compared to those in the control (Sham-treated) group. Continuous variables will be summarized descriptively (sample size, mean, standard deviation and error, minimum and maximum). Discrete variables will be summarized by frequency or percentage. All efficacy analyses will be based on the ITT Population. All

efficacy variables will be presented by 3.0 x 10<sup>6</sup> cells, 6.0 x 10<sup>6</sup> cells, and Sham treatments used for summary statistics.

For the endpoints with repeated post-baseline measures, the mean change from baseline in the efficacy parameters will be analyzed using a linear model accounting for repeated measures. The model will include main effects for treatment group, visit and treatment by visit interaction. The corresponding baseline parameter will be included as a covariate as well. Unless stated otherwise, the following visits will be used in the model: month 3, month 6, month 9 and month 12. An unstructured covariance model will be used. Treatment comparisons will be based on the modeled change from basline to month 3, month 6, month 9 and month 12. Primary end point for all efficacy analysis is at 12 months.

Post-baseline values that are missing will be imputed for each efficacy test using the Markov Chain Monte Carlo (MCMC) method. Ten copies of the dataset with a monotonic missing pattern will be genereated using the monotone data augmentaion method<sup>1, 2</sup> to impute the amount of missing data that is required to make the missing data pattern monotone before applying the multiple imputation algorithm. This method uses a non-informative Jefferys prior to derive the posterior mode from the expectation-maximization algorithm as starting values for the MCMC method. For each of the 10 monotonic missing pattern datasets, an additional 10 datasets will be imputed to replace missing values at scheduled visits for a total of 100 datasets. These datasets will be generated using a regression-based multiple imputation model.<sup>3</sup> For subjects with complete data up to a particular visit, a multiple regression model will be fit that includes the outcome at that visit as the dependent variable and outcomes at previous visits and treatment group as independent variables. Using these regression models, a missing value for a subject at a particular visit will be imputed as a draw from the predictive distribution given the outcomes at previous visits (some possibly imputed) and treatment group.<sup>3</sup>

The SAS MI procedure (ie PROC MI) using the monotone regression method will be used. The ROUND option will be used to round the imputed values to the same precision as the observed values and the minimum value for imputed will be specified as zero to avoid negative values. When an intended imputed value is less than the minimum, PROC MI will redraw another value for imputation. The linear model for repeated measures analyses will be performed separately for each of the 100 complete analysis data sets, and the results will be combined into one multiple imputation inference (estimated treatment effect and associated confidence interval and p-value)<sup>3, 4</sup> using PROC MIANLALYZE.

## 9.1 Best Corrected Visual Acuity (BCVA)

For BCVA, summary statistics of the total number of letters correct will be generated at each time point for 3 x  $10^6$  jCell dose, 6 x  $10^6$  jCell and Sham. Separate tables will be created for the Study Eye and the Non-Study Eye. In addition, change from baseline will also be summarized for each post baseline time point. For subjects who do not have a number score e.g. counting fingers (CF), hand motions (HM) or no light perception (NLP), letters missed will be considered to be 100 and letters correct will therefore be zero. The proportion of treated eyes with  $\geq 5$ ,  $\geq 10$  and  $\geq 15$  letter improvements at Month 3, Month 6, Month 9, Month 12 or Early Termination timepoints in both study eye and untreated eyes will be summarized. A global Chi-square test will be used for testing for any differences among treatment groups at Month 12. If the global test is significant at alpha equals 0.05, pairwise comparisions will be evaluated.

In addition, change in BCVA from baseline will be summarized for each dose level at Day 1, Day 7, Day 28, month 3, 6, 9, and 12 or Early Termination in both study eye and non-study eye for experimental J-cell groups and sham group. Each letter on EVA or ETDRS charts are equal to 0.02 logMar with starting reference for 20/20 is 0.0 LogMar, 20/200 is 1.0 logMar, and 20/1000 is 1.7 logMar. Conversion of ETDRS values to logMars are included in the following table:

| Letter Score | LogMAR Value | Snellen Equivalent |
|--------------|--------------|--------------------|
| 5 | 1.6 | 20/800 |
| 10 | 1.5 | 20/640 |
| 15 | 1.4 | 20/500 |
| 20 | 1.3 | 20/400 |
| 25 | 1.2 | 20/320 |
| 30 | 1.1 | 20/250 |
| 35 | 1.0 | 20/200 |
| 40 | 0.9 | 20/160 |
| 45 | 0.8 | 20/125 |
| 50 | 0.7 | 20/100 |
| 55 | 0.6 | 20/80 |
| 60 | 0.5 | 20/63 |
| 65 | 0.4 | 20/50 |
| 70 | 0.3 | 20/40 |
| 75 | 0.2 | 20/32 |
| 80 | 0.1 | 20/25 |
| 85 | 0.0 | 20/20 |
| 90 | -0.1 | 20/15 |
| 95 | -0.2 | 20/12 |

LogMAR = logarithm of the minimal angle of resolution.

Mean change in number of letters correct will be compared for the study eyes between each experimental j-cell group and control group at month 3, 6, 9 and 12 using the linear model specified in Section 9. LogMar scores and number of letters correct will be presented for table summaries, for mean changes LogMar and number of letters correct will be presented.

All subjects should have a measurable baseline BCVA value for the study based on the inclusion critieria. Subjects who cannot perform a BCVA assessment post-baseline are considered to have 0 letters correct, but are close to missing at random when the visit does not occur. The primary approach to post-baseline missing values for BCVA will be to consider records where a subject could not complete the assessment with 0 but in the case that no visit or an assessment was marked as not done, the recorded values will remain missing. The secondary approach will use Multiple Imputation to impute missing values as discussed in section 8.3.

Additionally, a sensitivity analysis modeling BCVA counts with a Poisson distribution may be considered if there is concern of severe departure from Guassian behavior.

## 9.2 Visual Field Examination

VF will be summarized for both study and non-study eye at specified time points. From the visual field examination, each area of vision will be added together using the V4e test target. The total area per eye will be compared at baseline, 6 months and 12 months using linear model specified in section 9. In the situation where kinetic visual fields are within 25% of normal ranges (>10,000 deg2), the III4e target size will be used in order to avoid a ceiling effect in subjects with near-normal V4e perimetry.

Subjects who can't perform kinetic field testing at baseline will be considered to have the lowest minimum measurable area of 6.8 square degrees. This value was obtained by using the smallest field area of any subject in the study using the V4e target.

Fixation capability proportions for both study eye and non-study eye will be summarized for each dose level at baseline, month 6, and 12 or Early Termination for experimental Jcell group and sham group. In addition, mean change in total field area will be summarized for the study eyes from baseline to month 6 and month 12 between each experimental j-cell group and control group using the linear model specified in Section 9. The primary approach for this analysis is to include subjects in the mITT population, which excludes patients with missing baseline values or who are unable to perform the assessment at baseline. Subjects who cannot perform a kinetic field assessment postbaseline are considered to have 6.8 square degrees but are close to missing at random when the visit does not occur. The secondary approach will be similar to primary approach and will use Multiple Imputation as discussed in section 8.3 for missing postbaseline visits. For the EE population, in the event that a baseline or post-baseline assessment could not be completed (inability to complete the test), the LOD will be used. Missing post-baseline values will be imputed using Multiple Imputation (see section 8.3). Subjects with completely missing baseline values (e.g. no visit or assessment attempted) will be considered inevaluable for this analysis.

## 9.3 Mobility

Mobility will be summarized for both study eye and non-study eye at specified time points. Descriptive statistics will be presented for Maximum step speed (MSS) and Critical illumination level (CIL) at baseline, month 6 and month 12. CIL is represented in even factor of 2 steps in the unit lux (e.g., 2 lux, 4 lux, 8 lux). MSS is a continuous variable. CIL scores will be converted to a scale score of -1 (cannot pass at the brightest

light level) to 13 (does not slow even with room lights off) and change in score from baseline and at each post baseline visit will be calculated. Conversion of CIL lux values to scale scores are included in the following table:

| CIL<br>(Lux) | Lights<br>off | 0.12 | 0.25 | 0.5 | 1.0 | 2.0 | 4.0 | 8.0 | 16 | 32 | 63 | 125 | 250 | 500 | No<br>Pass |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Scale<br>Score | 13 | 12 | 11 | 10 | 9 | 8 | 7 | 6 | 5 | 4 | 3 | 2 | 1 | 0 | -1 |

Mean changes from baseline in mobility test scores (CIL and MSS) will be compared in the study eyes between each experimental j-cell group and control group from baseline to month 6 and month 12 using the linear model specified in Section 9. Converted CIL scores and actual scores will be presented in listings and for table summaries, converted scores and actual scores will be presented. For mean changes converted scores will be presented.

Subjects who cannot perform mobility testing at baseline will be considered to have a passing lux level of 1000 or an equivalent scale score of -1 for CIL and 0 for MSS. This CIL scale value is proposed based on a similar recently FDA accepted test of low luminance mobility (the MLMT) and is analogous to using 0 letters correct on BCVA on subjects who have worse acuity than the test can assess.

The primary approach for this analysis is to include subjects in the mITT population, which excludes patients with missing or who cannot perform the test at baseline. Subjects who cannot perform a mobility assessment post-baseline are considered to have a -1 score for CIL and 0 value for MSS but are considered missing at random when the visit does not occur. The secondary approach is same as primry approach, except that when there is no visit or an assessment was marked as not done post-baseline, the recorded values will be imputed using Multiple Imputation as discussed in section 8.3. For the EE population, in the event that a baseline or post-baseline assessment has been attempted but subject could not perform the test, the LOD will be used at baseline and post-baseline. Missing post-baseline values will be imputed using Multiple Imputation. Subjects with completely missing baseline values (e.g. no visit or assessment attempted) will be considered inevaluable for this analysis.

## 9.4 Contrast Sensitivity (CS)

Contrast sensitivity will be summarized for both study eye and non-study eye at baseline, month 6 and month 12 with descriptive statistics for spatial frequency of 0.25, 0.5, 1.0,

2.0, 4.0, 8.0, and 12.0. For any spatial frequency with more than one threshold value (or trial), the values will be averaged (mean), and the single mean value for that spatial frequency will be reported. A single value indicates exploratory testing and does not represent repeatable trials and will not be analyzed. Mean change from baseline to month 6 and month 12 in CS thresholds for up to three spatial frequencies will be compared in the study eyes between each experimental j-cell group and control group from baseline to month 6 and month 12 using the linear model specified in Section 9.

The primary approach for this analysis is to include subjects in mITT population, which

excludes patients with missing baseline values or who could not perform the assessment at baseline (below LOD). Subjects who undergo CS assessments but do not have a value recorded post-baseline are assumed to be below the detection level of the instrument and therefore the lowest value detectable from other subjects will be used to replace the missing values. The contrast sensitivity value for spatial frequencies most commonly detected (0.5, 1.0, and 2.0 cycles per degree) is 1.28 indicating the subject can only see the target with the highest contrast possible. Values for subjects who do not have a visit record at all post-baseline are considered to be close to missing at random (visit missed or assessment not attempted) The secondary approach will be same as primary approach except that in the case that no visit or an assessment was marked as not done, the recorded values will be imputed using Multiple Imputations as discussed in section 8.3. For the EE population, in the event that a baseline or post-baseline assessment has been attempted but subject could not complete the test, the value will be considered to be the LOD. Missing post-baseline values will be imputed using Multiple Imputations. Subjects with completely missing baseline values (e.g. no visit or assessment attempted) will be considered inevaluable for this analysis.

## 9.5 Low Vision Visual Functional Questionnaire (LV-VFQ 48)

Low vision visual functional questionnaire overall scores and individual scale scores will be summarized for each subject at baseline, month 6 and month 12 with descriptive statistics (i.e., visual ability, reading, mobility, visual information, and visual motor).

The individual scale score (i.e., visual ability, reading, mobility, visual information, visual motor) mean changes from baseline to month 6 and month 12 in VA LV VFQ-48 will be summarized and compared between each experimental j-cell group and control group will be analyzed using repeated measurements specified in section 9 with a linear model for individual scale scores. For this analysis, all subjects can perform an individual score assessment, but will be considered close to missing at random when the visit does not occur. Therefore, in the case that this assessment was marked as not done at baseline, the subject will be considered inevaluable for this analysis. Where a post-

baseline value is missing, the approach will be to use Multiple Imputations as discussed in section 8.3.

## 10. SAFETY ANALYSES

All safety analyses will be based on the Safety population. Adverse events will be monitored by the investigator and the subject. The safety analyses of laboratory parameters will include descriptive statistics and AEs will include frequency counts and percentages. Summaries of AEs will be generated by type (AE or SAE), body system and preferred term, severity, and relationship to study product.

## 10.1 Study Drug Administration

Treatment compliance will be assessed via direct observation by the study investigator who is responsible for study drug administration. The cell dose and exact time of injection for test subjects will be recorded and the exact time of Sham injection for the control subjects will be recorded. Study drug administration responses will be tabulated for each treatment according to questions asked in the CRF, including whether the total dose was administered, whether there were any dose interruptions, whether there were any AEs observed, whether the subject's vital signs are comparable to pre-treatment of study drug injection, the subject was prescribed topical treatment after treatment of study drug injection.

#### 10.2 Adverse Events

All adverse event summaries will be restricted to Treatment Emergent Adverse Events (TEAE), which are defined as those AEs that occurred after dosing and those existing AEs that worsened during the study. If it cannot be determined whether the AE is treatment emergent due to a partial onset date then it will be counted as such. Verbatim terms on case report forms will be mapped to preferred terms and System Organ Classes using the Medical Dictionary for Regulatory Activities (MedDRA) (version 20.0).

Each adverse event summary will be displayed by treatment group. Summaries that are displayed by system organ class and preferred terms will be ordered by descending order of incidence of system organ class and preferred term within each system organ class. Summaries of the following types will be presented:

• Subject and event incidence of TEAEs by MedDRA system organ class and preferred term.

- Subject incidence of TEAEs by MedDRA system organ class, preferred term, and highest severity. At each level of subject summarization a subject is classified according to the highest severity if the subject reported more than one of the same event. Categories of severity will be "Mild", "Moderate", "Severe" and "Life Threatening" in this summary. The "Life Threatening" column will only be shown if at least 1 life-threatening AE is reported. If any AEs are reported with missing severity, then a footnote will be added to indicate how many AEs with missing severity were reported.
- Subject and event incidence of related TEAEs by MedDRA system organ class and preferred term. Related AEs are those reported as "Related", "Possibly Related" or relationship was not reported. At each level of subject summarization a subject is classified according to the closest relationship if the subject reported more than one event. AEs with a missing relationship will be considered related for this summary.
- Subject and event incidence of serious TEAEs by MedDRA system organ class and preferred term.

## 10.3 Clinical Laboratory Evaluation

Hematology and chemistry laboratory parameters will be summarized using descriptive statistics at baseline, day 28, month 3, month 6, and month 12 or early termination. Change from baseline in the laboratory parameters will also be presented, the baseline is defined as the last non-missing value recorded prior to the first dose of study drug.

Coagulation, infectious disease assessment (Hepatitis B and c, HIV lab test), PRA and DRA antibody test, and HLA typing results will be provided in a data listing.

No concerns are expected regarding the drug for laboratory results since the drug is expected to stay in the eye. As a result, no analysis using high/low flags will be carried out.

Urinalysis results will not be summarized but will be provided in data listing.

Separate listing of abnormal clinically significant lab values will be presented.

## 10.4 Vital Signs

Vital signs (systolic BP, diastolic BP, heart rate, respiration, temperature, and weight) will be summarized using descriptive statistics at baseline and at each post-baseline time

point. Changes from baseline will also be summarized. The baseline is defined as the last non-missing value recorded prior to the first dose of study drug.

## 10.5 Physical Examination

Physical examination results will be included in data listings only.

## 10.6 Ophthalmic AEs

## 10.6.1 Slit Lamp and Fundus Photography

Slit Lamp and Fundus Photography - The slit lamp exam will be summarized by eye structure. For eye structures of eyelids, eyelashes, conjunctiva, sclera, cornea, and iris, subjects will be tabulated by the categories of Normal, Abnormal NCS, and Abnormal CS at each time point, and percentages will be displayed. For anterior chamber flare, subjects will be tabulated by the flare grade and the categories of Abnormal NCS and Abnormal CS. For lens status, subjects will be tabulated as aphakic, pseudophakic, and phakic. For cataract type, subjects will be tabulated as nuclear, cortical, posterior sub capsular, and not applicable. Subjects will also be tabulated by grades of 1+, 2+, 3+ and 4+. For the fundus photography, results will be included in data listing only.

## 10.6.2 Intraocular Pressure (IOP)

IOP - Intraocular pressure and change in intraocular pressure will be summarized descriptively by time point.

#### 10.6.3 B-scan

B-scan results will be tabulated by Normal and Abnormal results at each time point and overall results will be counted as good or poor. B-scan results will also be tabulated by whether injected cells were visualized.

## **10.6.4 Dilated Fundoscopic Examination**

Dilated Fundoscopic Examination- for the vitreous exam, optic nerve exam, macula exam, and peripheral retina exam, counts and percentages of Normal, Abnormal NCS and Abnormal CS will be presented by eye and time point. When available, summaries of Severity (Mild +1, Moderate +2, Severe +3, Very Severe +4) will also be included.

## 10.6.5 Post Injection Clinical Vitreous Exam

Post Injection Clinical Vitreous Exam, counts and percentages will be summarized for method used (indirect ophthalmoscopy, fundus exam, slit lamp exam and other) and observations (cells, clumps, opacity, debris, strands, inflammation and other).

## **10.6.6 Optical Coherence Tomography (OCT)**

OCT results will be summarized in a table showing the counts and percentages of subjects whose eyes (both study eye and non-study eye) show cystoid macular edema present, and of those who do, how many cases involve the foveal center; epiretinal membrane formation present, and how many have evidence of retinal traction present.

#### 10.7.7 Autofluorescence

Fundus auto fluorescence will be summarized for both study eye and non-study eye at each time point with counts and incidence rates for each of the possible options of Normal, Abnormal NCS, and Abnormal CS.

#### 11. REFERENCES

- 1. Li KH (1988) Imputation using Markov chains. J Statist Comp Simul; 30:57-79.
- 2. Liu C (1993) Bartlett's decomposition of the posterior distribution of the covariance for normal monotone ignorable missing data. J Mult Anal; 46:198-206.
- 3. Little R, Yau L (1996) Intent-to-treat analysis for longitudinal studies with drop-outs. Biometrics; 52:1324-1333.
- 4. Schafer, JL (1997) Analysis of Incomplete Multivariate Data, New York: Chapman and Hall.
- 5. <a href="http://www.rand.org/content/dam/rand/www/external/health/surveys\_tools/vfq/vfq25">http://www.rand.org/content/dam/rand/www/external/health/surveys\_tools/vfq/vfq25</a> <a href="maintaile-maintail
- 6. Mangione, CM, Lee PP, Gutierrez, PR, et al. Development of the 25-item National Eye Institute Visual Function Questionnaire (VFQ-25). Archives of Ophthalmology, 2001. 119: 1050-1058
- 7. <a href="http://eva.jaeb.org/test">http://eva.jaeb.org/test</a> information/Algorithm EETDRS.pdf

#### **APPENDICES**

## Appendix A: Presentation of Data and Programming Specifications

#### General

- Specialized text styles, such as bold, italics, borders, shading, superscripted and subscripted text will not be used in tables and data listings unless they add significant value to the table, figure, or data listing.
- Only standard keyboard characters are to be used in tables and data listings.
- Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used on a table or data listing.
- Hexadecimal character representations are allowed (e.g.,  $\mu$ , a,  $\beta$ ).
- All footnotes will be left justified and at the bottom of a page. Footnotes should be used sparingly and must add value to the table or data listing.

#### **Tables**

- Formal organization of tabulations may be changed during programming if appropriate, e.g., tables for the different variables may be combined into a single table, or tables with more than one variable may be split into several tables.
- Means and medians will be presented to one more decimal place than the raw data. Standard deviations will be presented to two more decimal places than the raw data. Minimums and maximums will be reported with the same number of decimal places as the raw data.
- Percentages will be presented to the tenths place.
- For frequency counts of categorical variables, categories with zero counts will not be displayed.

#### Listings

- Formal organization of the listing may be changed during programming if appropriate, e.g., additional variables may be included, change in the column order, or the listing may be split into multiple parts due to space constraints, etc.
- If not otherwise specified, all data listings will be sorted by sequence/treatment, center, subject number, visit, and date/time as appropriate.
- All date values will be presented in an ISO8601 date (e.g., 2018-10-11) format.

• All observed time values will be presented using a 24-hour clock HH:MM:SS format (e.g., 01:35:45 or 11:26). Seconds will only be reported if they were measured as part of the study.

## Missing or incomplete dates (i.e., AEs and concomitant medications)

The most conservative approach will be systematically considered. If the AE onset date is missing / incomplete, it is assumed to have occurred during the study treatment phase (i.e., considered a TEAE) except if the partial onset date or other data such as the stop date, indicates differently. Similarly, a medication with partial start and stop dates could be considered as both a prior and concomitant treatment.

The following algorithms will be applied to missing and incomplete start and stop dates:

## **Start Dates**

- If the day portion of the start date is missing, then the start date will be estimated to be equal to the date of first dose of study drug, provided the start month and year are the same as the first dose of study drug and the stop date is either after the first dose of study drug or completely missing. Otherwise, the missing day portion will be estimated as '01'.
- If both the day and month portions of the start date are missing, then the start date will be estimated to be equal to the date of first dose of study drug, provided the start year is the same as the first dose of study drug and the stop date is either after the first dose of study drug or completely missing. Otherwise, the event will be assumed to start on the first day of the given year (e.g., ??-???-2013 is estimated as 01-JAN-2013).
- If the start date is completely missing and the stop date is either after the dose of study drug or completely missing, the start date will be estimated to be the day of study drug dosing. Otherwise, the start date will be estimated to be the first day of the same year as the stop date. All other non-AE and non-concomitant medication day calculations where only partial dates are available will be handled as follows: the first day of the month will be used in the calculations if the day part of a start date is missing while January 1 will be employed if both the month and day parts of a start date are missing.

#### **Stop Dates**

• If only the day of resolution is unknown, the day will be assumed to the last of the month (e.g., ??-JAN-2013 will be treated as 31-JAN-2013).

- If both the day and month of resolution are unknown, the event will be assumed to have ceased on the last day of the year (e.g., ??-???-2013 will be treated as 31-DEC-2013).
- If the stop date is completely missing or the event is continuing, the event will be assumed to be after first dose of study drug and will be imputed using the last known date on the study.

## Appendix B: List of Tables, Figures, and Listings

The following TLF numbering is completed according to ICH E3 guidelines. The ICH heading number and description are in **bold**. Minor changes from this planned index do not need to be amended in the SAP.

Formal organization of tabulations may be changed during programming if appropriate, e.g., tables for the different variables may be combined into a single table, or tables with more than one variable may be split into several tables.

## **List of Tables**

| ICH | Table | |
|---|---|---|
| Heading | Number | Table Description |
| 14.1 | | DEMOGRAPHIC DATA |
| | 14.1.1 | Subject Disposition |
| | 14.1.2 | Demographic and Baseline Characteristics (Safety/ITT |
| | | Population) |
| 14.2 | | EFFICACY DATA |
| | 14.2.1.1 | Best Corrected Visual Acuity (ETDRS): Study Eye Number |
| | | of Letters Correct (ITT Population) |
| | 14.2.1.2 | Best Corrected Visual Acuity (ETDRS): Non-Study Eye |
| | | Number of Letters Correct (ITT Population) |
| | 14.2.1.3 | Categorical Analysis of Best Corrected Visual Acuity |
| | | (ETDRS): Study Eye Number of Letters Correct (ITT |
| | | Population) |
| | 14.2.1.4 | Categorical Analysis of Best Corrected Visual Acuity |
| | | (ETDRS): Non-Study Eye Number of Letters Correct (ITT |
| | | Population) |
| | 14.2.1.5.1 | Mean Change in Best Corrected Visual Acuity (ETDRS): |
| | | Study Eye Number of Letters Correct (ITT Population) |
| | 14.2.1.5.2 | Mean Change in Best Corrected Visual Acuity (ETDRS): |
| | | Study Eye Number of Letters Correct using Multiple |
| | | Imputation (ITT Population) |
| | 14.2.1.5.3 | Mean Change in Best Corrected Visual Acuity (FrACT): |
| | | Study Eye LogMar Scores (ITT Population) |

| ICH | Table | |
|---|---|---|
| Heading | Number | Table Description |
| | 14.2.1.5.4 | Mean Change in Best Corrected Visual Acuity (FrACT): |
| | | Study Eye LogMar Scores using Multiple Imputation (ITT |
| | | Population) |
| | 14.2.2.1 | Visual Field :Study Eye (ITT Population) |
| | 14.2.2.2 | Visual Field: Non-Study Eye (ITT Population) |
| | 14.2.2.3.1 | Mean Change in Visual Field: Study Eye (mITT Population) |
| | 14.2.2.3.2 | Mean Change in Visual Field: Study Eye using Multiple |
| | | Imputation (mITT Population) |
| | 14.2.2.3.3 | Mean Change in Visual Field: Study Eye (EE Population) |
| | 14.2.3.1 | Mobility: Study Eye (ITT population) |
| | 14.2.3.2 | Mobility: Non-Study Eye (ITT Population) |
| | 14.2.3.3.1 | Mean Change in Mobility: Study Eye (mITT Population) |
| | 14.2.3.3.2 | Mean Change in Mobility: Study Eye using Multiple |
| | | Imputation (mITT Population) |
| | 14.2.3.3.3 | Mean Change in Mobility: Study Eye (EE Population) |
| | 14.2.4.1 | Contrast Sensitivity: Study Eye (ITT Population) |
| | 14.2.4.2 | Contrast Sensitivity: Non-Study Eye (ITT Population) |
| | 14.2.4.3.1 | Mean Change in Contrast Sensitivity: Study Eye (mITT |
| | | Population) |
| | 14.2.4.3.2 | Mean Change in Contrast Sensitivity: Study Eye using |
| | | Multiple Imputation (mITT Population) |
| | 14.2.4.3.3 | Mean Change in Contrast Sensitivity: Study Eye (EE |
| | | Population) |
| | 14.2.5.1.1 | Mean Change in Low Vision Functional Questionnaire: |
| | | Person (mITT Population) |
| | 14.2.5.1.2 | Mean Change in Low Vision Functional Questionnaire: |
| | | Person using Multiple Imputation (mITT Population) |
| 110 | | |
| 14.3 | | SAFETY DATA |
| | 14.3.1 | Study Drug Administration (Safety Population) |
| 14.3.1 | | Displays of Adverse Events |
| | 14.3.1.1 | TEAEs by System Organ Class and Preferred Term (Safety |
| | 44045 | Population) |
| | 14.3.1.2 TEAEs by System Organ Class, Preferred Term and | |
| | | Maximum Severity (Safety Population) |

| ICH | Table | |
|---|---|---|
| Heading | Number | Table Description |
| | 14.3.1.3 | Related to Study Drug TEAEs by System Organ Class and |
| | | Preferred Term (Safety Population) |
| | 14.3.1.4 | Serious TEAEs by System Organ Class and Preferred Term |
| | | (Safety Population) |
| | 14.3.4.1 | Hematology (Safety Population) |
| | 14.3.4.2 | Chemistry (Safety Population) |
| | 14.3.4.3 | Vital Signs (Safety Population) |
| | 14.3.4.4.1 | Slit Lamp Examination: Study Eye (Safety Population) |
| | 14.3.4.4.2 | Slit Lamp Examination: Non-Study Eye (Safety Population) |
| | 14.3.4.5.1 | Intraocular Pressure (IOP): Study Eye (Safety Population) |
| | 14.3.4.5.2 | Intraocular Pressure (IOP): Non-Study Eye (Safety |
| | | Population) |
| | 14.3.4.6.1 | B-Scan Study Eye (Safety Population) |
| | 14.3.4.6.2 | B-Scan: Non-Study Eye (Safety Population) |
| | 14.3.4.7.1 | Dilated Fundoscopic Examination: Study Eye (Safety |
| | | Population) |
| | 14.3.4.7.2 | Dilated Fundoscopic Examination: Non-Study Eye (Safety |
| | | Population) |
| | 14.3.4.8 | Post Injection Clinical Vitreous Exam: Study Eye (Safety |
| | | Population) |
| | 14.3.4.9.1 | Optical Coherence Tomography (OCT): Study Eye, |
| | | Categorical Analysis (Safety Population) |
| | 14.3.4.9.2 | Optical Coherence Tomography (OCT): Non-Study Eye, |
| | | Categorical Analysis (Safety Population) |
| | 14.3.4.10.1 | Autofluorescence: Study Eye (Safety Population) |
| | 14.3.4.10.2 | Autofluorescence: Non-Study Eye (Safety Population) |

# **List of Data Listings**

| ICH | Listing | |
|---|---|---|
| Heading | Number | Listing Description |
| 16.2.1 | 16.2.1.1 | Subject Disposition (All Subjects) |
| 16.2.2 | 16.2.2.1 | Protocol Deviations (All Subjects) |
| | 16.2.2.2 | Inclusion/Exclusion Criteria (All Subjects) |
| 16.2.4 | 16.2.4.1 | Demographics and Baseline Characteristics (Safety |
| | | Population) |
| | 16.2.4.2 | Medical History (Safety Population) |
| | 16.2.4.3 | Ocular Medical History (Safety Population) |
| 16.2.5 | 16.2.5 | Study Drug Administration (Safety Population) |
| 16.2.6 | 16.2.6.1 | Best Corrected Visual Acuity (ETDRS and/or FrACT) |
| | | (ITT Population) |
| | 16.2.6.2 | Optical Coherence Tomography (OCT) (Safety |
| | | Population) |
| | 16.2.6.3 | Autofluorescence (Safety Population) |
| | 16.2.6.4 | Visual Field Examination (ITT Population) |
| | 16.2.6.5 | Mobility (ITT Population) |
| | 16.2.6.6 | Contrast Sensitivity (ITT Population) |
| | 16.2.6.7 | Low Vision Functional Questionnaire (LV-VFQ28) (ITT |
| | | Population) |
| 16.2.7 | 16.2.7.1 | Adverse Events (Safety Population) |
| | 16.2.7.2 | Serious Adverse Events (Safety Population) |
| | 16.2.7.3 | Related Adverse Events (Safety Population) |
| | 16.2.7.4 | Post Injection Clinical Vitreous Exam (Safety Population) |
| 16.2.8 | 16.2.8.1 | Hematology (Safety Population) |
| | 16.2.8.2 | Chemistry (Safety Population) |
| | 16.2.8.3 | Urinalysis/Microscopic Exam (Safety Population) |
| | 16.2.8.4 | Clinically Significant Lab Values(Safety Population) |
| | 16.2.8.5 | Coagulation Function (Safety Population) |
| | 16.2.8.6 | Infectious Disease Assessments (Safety Population) |
| | 16.2.8.7 | HLA Typing (Safety Population) |
| | 16.2.8.8 | Vital Signs (Safety Population) |
| | 16.2.8.9 | Physical Examination (Safety Population) |
| | 16.2.8.10 | Prior and Concomitant Medications (Safety Population) |
| | 16.2.8.11 | Pregnancy Test (Safety Population) |

| ICH | Listing | |
|---------|-------------|-----------------------------------------------------|
| Heading | Number | Listing Description |
| | 16.2.8.12 | PRA and DRA Antibody Test Results (Safety |
| | | Population) |
| | 16.2.8.13.1 | Slit Lamp (OD) (Safety Population) |
| | 16.2.8.13.2 | Slit Lamp (OS) (Safety Population) |
| | 16.2.8.14 | Intraocular Pressure (IOP) (Safety Population) |
| | 16.2.8.15 | B-Scan (Safety Population) |
| | 16.2.8.16 | Dilated Fundoscopic Examination (Safety Population) |
| | 16.2.8.17 | Fundus Photographs (Safety Population) |

**Appendix C: Table Layouts** 

jCyte, Inc. Page 1 of x Protocol: JC-02

**Table 14.1.1 Subject Disposition** All Enrolled Subjects

| | Sham | 3.0 x 10 <sup>6</sup> hRPC | 6.0 x 10 <sup>6</sup> hRPC | Total |
|---|---|---|---|---|
| Subjects Enrolled | N | N | N | N |
| ITT Population [1] | n (%) | n (%) | n (%) | n (%) |
| Safety Population [2] | n (%) | n (%) | n (%) | n (%) |
| Primary Reason for Discontinuation | | | | |
| Completed Study | n (%) | n (%) | n (%) | n (%) |
| Adverse Event | n (%) | n (%) | n (%) | n (%) |
| Lack of Efficacy | n (%) | n (%) | n (%) | n (%) |
| Lost to Follow Up | n (%) | n (%) | n (%) | n (%) |
| Non-Compliance with Study Treatment | n (%) | n (%) | n (%) | n (%) |
| Physician Decision | n (%) | n (%) | n (%) | n (%) |
| Pregnancy | n (%) | n (%) | n (%) | n (%) |
| Progressive Disease | n (%) | n (%) | n (%) | n (%) |
| Protocol Deviation | n (%) | n (%) | n (%) | n (%) |
| Recovery | n (%) | n (%) | n (%) | n (%) |
| Study Terminated by Sponsor | n (%) | n (%) | n (%) | n (%) |
| Withdrawn by Subject | n (%) | n (%) | n (%) | n (%) |
| Death | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) |

Note: Percentages based on Subjects Enrolled.

path\t program.sas date

Programmer Note: only shows primary reason for Discontinuation that has results.

Programmer Note: If any of the rows in primary reason for Discontinuation shows 0 frequencies drop that row. Same for all frequency tables.

<sup>[1]</sup> All randomized subjects who provide any post-randomization data. [2] Received any amount of study treatment (including sham).

Page 1 of x jCyte, Inc. Protocol: JC-02

**Table 14.1.2 Demographic and Baseline Characteristics** Safety/ITT Population

| | Sham<br>(N=) | $3.0 \times 10^6 \text{ hRPC}$ (N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| Age (years) [1] | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx x (xx x) | xx x (xx x) |
| Median | XX X | XX X | XX X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Sex | | | |
| Male | n (%) | n (%) | n (%) |
| Female | n (%) | n (%) | n (%) |
| Ethnicity | | | |
| Hispanic or Latino | n (%) | n (%) | n (%) |
| Not Hispanic or Latino | n (%) | n (%) | n (%) |
| Race | | | |
| American Indian or Alaska Native | n (%) | n (%) | n (%) |
| Asian | n (%) | n (%) | n (%) |
| Black or African American | n (%) | n (%) | n (%) |
| Native Hawaiian or Other Pacific Islander | n (%) | n (%) | n (%) |
| White | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) |
| Multiple Races Checked | n (%) | n (%) | n (%) |

<sup>[1]</sup> Age determined by comparing date of birth to date of informed consent.
[2] Baseline is defined as the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date time
**Table 14.1.2 Demographics and Baseline Characteristics** Safety/ITT Population

| | Sham | $3.0 \times 10^6 hRPC$ | 6.0 x 10 <sup>6</sup> hRPC |
|---|---|---|---|
| | (N=) | (N=) | (N=) |
| Study Eye | | | |
| OD (Right) | n (%) | n (%) | n (%) |
| OS (Left) | n (%) | n (%) | n (%) |
| Height (cm) [2] | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | XX X | XX.X | XX.X |
| Min, Max | XX, XX | xx, xx | xx, xx |
| Weight (kg) [2] | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx.x(xx.x) |
| Median | xx x | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx |

Programmer note: For the subsequent tables, use Table 14.1.2 to determine which columns to include.

<sup>[1]</sup> Age determined by comparing date of birth to date of informed consent.
[2] Baseline is defined as the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date

jCyte, Inc. Page 1 of x

Protocol: JC-02

## **Table 14.2.1.1** Best Corrected Visual Acuity (ETDRS): Study Eye **Number of Letters correct** ITT Population

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| Baseline [1] | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | XX, XX | xx, xx | xx, xx |

| Day 1 | | | |
|-----------|-------------|-------------|-------------|
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | XX, XX | XX, XX | XX, XX |

<sup>[1]</sup> Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the value at the screening visit. path\t program.sas date time

Programmer Note: Continue table for VisitsDay 1, Day 7, Day 28, Month 3, Month 6, Month 9, Month 12 or Early Termination Programmer Note: Table 14.2.1.2 will contain the same information for the Non-Study Eye.

Programmer Note: Original values will be used and no thresh hold limit or imputed values used in this table.

jCyte, Inc. Page 1 of x

Protocol: JC-02

**Table 14.2.1.3** Categorical Analysis of Best Corrected Visual Acuity (ETDRS): Study Eye **Number of Letters correct** ITT Population

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) | Global Test [1] |
|---|---|---|---|---|
| Proportion of Subjects with Specified increase in letters correct for any Post<br>Baseline Assessment | (n=) | (n=) | (n=) | |
| >=5 Letters Increase | n (%) | n (%) | n (%) | |
| >=10 Letters Increase | n (%) | n (%) | n (%) | |
| >=15 Letters Increase | n (%) | n (%) | n (%) | |
| Proportion of Subjects with Specified increase in letters correct at Month 3 | (n=) | (n=) | (n=) | |
| >=5 Letters Increase | n (%) | n (%) | n (%) | |
| >=10 Letters Increase | n (%) | n (%) | n (%) | |
| >=15 Letters Increase | n (%) | n (%) | n (%) | |
| Proportion of Subjects with Specified increase in letters correct at Month 6 | (n=) | (n=) | (n=) | |
| >=5 Letters Increase | n (%) | n (%) | n (%) | |
| >=10 Letters Increase | n (%) | n (%) | n (%) | |
| >=15 Letters Increase | n (%) | n (%) | n (%) | |
| Proportion of Subjects with Specified increase in letters correct at Month 9 | (n=) | (n=) | (n=) | |
| >=5 Letters Increase | n (%) | n (%) | n (%) | |
| >=10 Letters Increase | n (%) | n (%) | n (%) | |
| >=15 Letters Increase | n (%) | n (%) | n (%) | |
| Proportion of Subjects with Specified increase in letters correct at Month 12 | (n=) | (n=) | (n=) | |
| >=5 Letters Increase | n (%) | n (%) | n (%) | X XXXX |
| P-value [2] | ` ′ | x.xxxx | x xxxx | |
| >=10 Letters Increase | n (%) | n (%) | n (%) | X XXXX |
| P-value [2] | | x.xxxx | x xxxx | |
| >=15 Letters Increase | n (%) | n (%) | n (%) | X XXXX |
| P-value [2] | | X.XXXX | x xxxx | |

ppath\t\_program.sas date time

<sup>[1]</sup> From chi-square tests any difference in any treatment groups.
[2] Pairwise chi-square tests for differences in control and treatment groups.

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that particular time point. Programmer Note: Table 14.2.1.4 will contain the same information for the Non-Study Eye Programmer Note: populate the [2] if the [1] is significant at alpha= 0.05. Programmer Note: Original values will be used and no thresh hold limit or imputed values used in this table.


Table 14.2.1.5.1
Mean Change in Best Corrected Visual Acuity (ETDRS): Study Eye
Number of Letters correct
ITT Population

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| Number of Letters Correct at Baseline <sup>[1]</sup> | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | xx x | xx.x | XX X |
| Min, Max | XX, XX | xx, xx | xx, xx |
| Number of Letters Correct at Month 3 , continue for Month 6 ar 9 | nd | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | xx x | xx.x | XX X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Change from Baseline to Month 3, continue for Month 6 and 9 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | xx x | xx.x | XX X |
| Min, Max | xx, xx | XX, XX | XX, XX |
| LS Mean (SE) <sup>[2]</sup> | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| LS Mean Difference [95%CI] (SE) [2] | , | xx x [xx x, xx.x] | xx x [xx x, xx x] |
| Number of Letters Correct at Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Change from Baseline to Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx x (xx x) |
| Median | XX X | xx.x | XX X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| LS Mean (SE) [2] | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| LS Mean Difference [95%CI] (SE) [2] | | xx x [xx x, xx.x] | xx x [xx x, xx x] |
| P-value <sup>[2]</sup> | | x.xxxx | X XXXX |

- [1] Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the value at the screening visit.
- [2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC Sham, 6.0 x 10<sup>6</sup> hRPC Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix.

  path\t program.sas date time

Programmer Note: Continue table for Visits: Month 3,6,9 and Month 12.

Programmer Note: Table 14.2.1.5.2 Mean Change in Best Corrected Visual Acuity (ETDRS): Study Eye Number of Letters Correct using Multiple Imputation (ITT Population) l

- [1] Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the value at the screening visit.
- [2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC Sham, 6.0 x 10<sup>6</sup> hRPC Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix. This model incorporates missing data using multiple imputation.

Programmer Note: Table 14.2.1.5.3 Mean Change in Best Corrected Visual Acuity (FrACT): Study Eye LogMar scores (ITT Population) l

- [1] Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the value at the screening visit.
- [2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC Sham, 6.0 x 10<sup>6</sup> hRPC Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix. This model incorporates missing data using multiple imputation

Programmer Note: Table 14.2.1.5.4 Mean Change in Best Corrected Visual Acuity (FrACT): Study Eye LogMar scores using Multiple Imputation (ITT Population) l

- [1] Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the value at the screening visit.
- [2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC Sham, 6.0 x 10<sup>6</sup> hRPC Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix. This model incorporates missing data using multiple imputation.

jCyte, Inc. Protocol: JC-02 Page 1 of x

**Table 14.2.2.1** Visual Field : Study Eye (cont.) ITT Population

| | Sham<br>(N=) | $3.0 \times 10^6 \text{ hRPC}$<br>(N=) | $6.0 \times 10^6 \text{ hRPC}$<br>(N=) |
|---|---|---|---|
| Fixation Stability | | . , | , , |
| Study Eye | | | |
| Baseline [1] | (n=) | (n=) | (n=) |
| 1=Unable to Find Fixation Target | n (%) | n (%) | n (%) |
| 2 = Able to Maintain Fixation 25% of the Time | n (%) | n (%) | n (%) |
| 3=Able to Maintain Fixation 50% of the Time | n (%) | n (%) | n (%) |
| 4 = Able to Maintain Fixation 75% of the Time | n (%) | n (%) | n (%) |
| 5=Able to Maintain Fixation 100% of the Time | n (%) | n (%) | n (%) |
| Continue for Month 6, and 12 | (n=) | (n=) | (n=) |
| 1=Unable to Find Fixation Target | n (%) | n (%) | n (%) |
| 2 = Able to Maintain Fixation 25% of the Time | n (%) | n (%) | n (%) |
| 3=Able to Maintain Fixation 50% of the Time | n (%) | n (%) | n (%) |
| 4 = Able to Maintain Fixation 75% of the Time | n (%) | n (%) | n (%) |
| 5=Able to Maintain Fixation 100% of the Time | n (%) | n (%) | n (%) |

<sup>[1]</sup> Baseline is defined as the value obtained at the baseline visit. path\t\_program.sas date time

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that particular time point... Programmer Note: Original values will be used and no thresh hold limit or imputed values used in this table.

## Table 14.2.2.1 Visual Field: Study Eye ITT Population

| | Sham<br>(N=) | $3.0 \times 10^6 \text{ hRPC}$ (N=) | $6.0 \times 10^6 \text{ hRPC}$<br>(N=) |
|---|---|---|---|
| | (11-) | (IV-) | (IN-) |
| Total Field Area | | | |
| Study Eye | | | |
| Baseline [1] | | | |
| n | | | |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| Total Field Area at Month 6 Continue for Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | XX, XX | xx, xx | XX, XX |

<sup>[1]</sup> Baseline is defined as the value obtained at the baseline visit.

path\t\_program.sas date time

*Programmer Note:* Field Area Total will be calculated by taking the sum of all the individual field areas (i.e., islands) for a subject with same visit, same eye, same date and time with same stimulus size. Only the stimulus size V4e is used and recorded in all subjects.

Field area total is same as adjusted calculated Size in CRF.

Programmer Note: Table 14.2.2.2 will contain the same information for the Non-Study Eye

Programmer Note: Total Visual Field area will be calculated using for a subject with same visit, same date and time with same stimulus size then sum all the adjusted calculate size and put the value in that visit.

If a subject has different Stimulus size use the following rule.

If stimulus size sum for V4e is >10,000 then use III4e stimulus size sum for total field area in visits. If at baseline stimulus size III4e is used same has to use for all other visits.

Programmer Note: Original values will be used and no thresh hold limit or imputed values used in this table.

Table 14.2.2.3.1 Mean Change in Visual Field: Study Eye mITT Population

| Total Visual Field Area at Baseline <sup>[1]</sup> n Mean (SD) Median Min, Max Total Visual Field Area at Month 6 | n<br>xx x (xx x)<br>xx x<br>xx, xx<br>n<br>xx x (xx x) | n<br>xx.x (xx.x)<br>xx.x<br>xx, xx | n<br>xx x (xx x)<br>xx x<br>xx, xx |
|---|---|---|---|
| n<br>Mean (SD)<br>Median<br>Min, Max | xx x (xx x) xx x xx, xx | xx.x (xx.x)<br>xx.x<br>xx, xx | xx x (xx x)<br>xx x |
| Mean (SD) Median Min, Max | xx x (xx x) xx x xx, xx | xx.x (xx.x)<br>xx.x<br>xx, xx | xx x (xx x)<br>xx x |
| Median<br>Min, Max | xx x<br>xx, xx | XX.X<br>XX, XX | XX X |
| Min, Max | xx, xx | xx, xx | |
| Total Visual Field Area at Month 6 | | n | |
| | | n | |
| n | xx x (xx x) | 11 | n |
| Mean (SD) | AA A (AA A) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | XX, XX | XX, XX | xx, xx |
| Change from Baseline to Month 6 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | XX, XX | xx, xx | XX, XX |
| LS Mean (SE) [2] | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| LS Mean Difference [95%CI] (SE) [2] | | xx x [xx x, xx.x] | xx x [xx x, xx x] |
| Total Visual Field Area at Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | XX, XX | xx, xx | xx, xx |
| Change from Baseline to at Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| LS Mean (SE) [2] | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| LS Mean Difference [95%CI] (SE) [2] | | xx x [xx x, xx.x] | xx x [xx x, xx x] |
| P-value <sup>[2]</sup> | | X.XXXX | x xxxx |

<sup>[1]</sup> Baseline is defined as the value obtained at the baseline visit.

[2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC – Sham, 6.0 x 10<sup>6</sup> hRPC – Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix.

path/t program.sas date time

Programmer Note: Continue table for Visits: Month 6, Month 12

Programmer Note: Total Visual Field area will be calculated using for a subject with same visit, same date and time with same stimulus size then sum all the adjusted calculate size and put the value in that visit.

If a subject has different Stimulus size use the following rule.

If stimulus size sum for V4e is > 10,000 then use III4e stimulus size sum for total field area in visits. If at baseline stimulus size III4e is used same has to use for all other visits.

Programmer Note: Table 14.2.2.3.2 Mean Change in Visual Field: Study Eye using Multiple Imputation (mITT Population)

- [1] Baseline is defined as the value obtained at the baseline visit.
- [2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC Sham, 6.0 x 10<sup>6</sup> hRPC Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix. This model incorporates missing data using multiple imputation

Programmer Note: Table 14.2.2.3.3 Mean Change in Visual Field: Study Eye (EE Population)

- [1] Baseline is defined as the value obtained at the baseline visit.
- [2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC Sham, 6.0 x 10<sup>6</sup> hRPC Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix.

Table 14.2.3.1 Mobility: Study Eye ITT Population

| | Sham<br>(N=) | $3.0 \times 10^6 \text{ hRPC}$ (N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| Maximum Step Speed | | | |
| Baseline [1] | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx x (xx x) | xx.x(xx.x) |
| Median | XX X | XX X | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Month 6 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx x (xx x) | xx.x(xx.x) |
| Median | XX X | xx x | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx x (xx x) | xx.x (xx.x) |
| Median | XX X | XX X | xx.x |
| Min, Max | XX, XX | xx, xx | XX, XX |

<sup>[1]</sup> Baseline is defined as the value obtained at the baseline visit. path\t program.sas date time

Programmer Note: Continue table for Visits: Month 6, Month 12... Also continue for Critical Illumination Level and converted Critical Illumination level (mean, SD, median, min and max). Use both original and converted scores for analysis...

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that particular time point.

Programmer Note: Table 14.2.3.2 will contain the same information for the Non-Study Eye

Programmer Note: no missing imputations or thresh hold values will be used in this table. Use original values.

Table 14.2.3.3.1 Mean Change in Mobility: Study Eye mITT Population

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| Maximum Step Speed at Baseline <sup>[1]</sup> | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Maximum Step Speed at Month 6 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| Change from Baseline to Month 6 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | xx x |
| Min, Max | XX, XX | xx, xx | XX, XX |
| LS Mean (SE) [2] | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| LS Mean Difference [95%CI] (SE) <sup>[2]</sup> | | xx x [xx x, xx.x] | xx x [xx x, xx x] |
| Maximum Step Speed at Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Change from Baseline to at Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | xx.x | XX X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| LS Mean (SE) [2] | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| LS Mean Difference [95%CI] (SE) <sup>[2]</sup> | | xx x [xx x, xx.x] | xx x [xx x, xx x] |
| P-value <sup>[2]</sup> | | X.XXXX | x xxxx |

<sup>[1]</sup> Baseline is defined as the value obtained at the baseline visit.

[2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC – Sham, 6.0 x 10<sup>6</sup> hRPC - Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix.

path\t program.sas date time

Programmer Note: Continue table for Critical Illumination for Visits: Month 6, Month 12. Also continue for Critical Illumination Level. Converted scores need to use for analysis.

Programmer Note: Table 14.2.3.3.2 Mean Change in Mobility: Study Eye using Multiple Imputation (mITT Population)

- [1] Baseline is defined as the value obtained at the baseline visit.
- [2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC Sham, 6.0 x 10<sup>6</sup> hRPC Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix. This model incorporates missing data using multiple imputation

Programmer Note: Table 14.2.3.3.3 Mean Change in Mobility: Study Eye (EE Population)

- [1] Baseline is defined as the value obtained at the baseline visit.
- [2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC Sham, 6.0 x 10<sup>6</sup> hRPC Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix.

Table 14.3.4.1 Contrast Sensitivity: Study Eye ITT Population

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | $6.0 \times 10^6 \text{ hRPC}$<br>(N=) |
|---|---|---|---|
| 0.25 | | | |
| 0.25 Baseline [1] | | | |
| | | _ | |
| n<br>M (GD) | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX X | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| Month 6 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX X | xx.x | xx.x |
| Min, Max | XX, XX | xx, xx | xx, xx |
| Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX X | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> Baseline is defined as the value obtained at the baseline visit. path\t program.sas date time

Programmer Note: Continue table for Visits: Month 6, Month 12. Also continue for 0.5 (20/1200), 1.0, 2.0, 4.0, 8.0, 12.0. Or all available visits and frequencies.

Programmer Note: take first OECS3 value and add it to all OETHRVAL and take mean of all those values. Use these means to calculate continuous variables. If only one value in OECS3 and no values in OETHRVAL, then ignore that value and do not include in calculating mean.

Programmer Note: Table 14.2.4...2 will contain the same information for the Non-Study Eye

Programmer Note: in this table use means with two are more data points. Don't use single values in mean calculation.

**Table 14.2.4.3.1** Mean Change in Contrast Sensitivity: Study Eye mITT Population

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| 0.5 Threshold CS Value at Baseline <sup>[1]</sup> | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | xx.x | XX X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| 0.5 Threshold CS Value at Month 6 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Change from Baseline to Month 6 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | xx.x | XX X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| LS Mean (SE) <sup>[2]</sup> | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| LS Mean Difference [95%CI] (SE) <sup>[2]</sup> | | xx x [xx x, xx.x] | xx x [xx x, xx x] |
| 0.5 Threshold CS Value at Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Change from Baseline to Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | xx.x | XX X |
| Min, Max | XX, XX | xx, xx | XX, XX |
| LS Mean (SE) <sup>[2]</sup> | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| LS Mean Difference [95%CI] (SE) <sup>[2]</sup> | | xx x [xx x, xx.x] | xx x [xx x, xx x] |
| P-value <sup>[2]</sup> | | x.xxxx | X XXXX |

<sup>[1]</sup> Baseline is defined as the value obtained at the baseline visit.

[2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC – Sham, 6.0 x 10<sup>6</sup> hRPC – Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix.

path\t program.sas date time

Programmer Note: Continue table for Visits: Month 6, Month 12. Also continue for 0.5 (20/1200), 1.0, 2.0, 4.0, 8.0, 12.0. Or all available visits and frequencies...

Programmer Note: take first OECS3 value and add it to all OETHRVAL and take mean of all those values. Use these means to calculate continuous variables. If only one value in OECS3 and no values in OETHRVAL, then ignore that value and do not include in calculating mean.

Programmer Note: Table 14.2.4.3.2 Mean Change in Contrast Sensitivity: Study Eye using Multiple Imputation (mITT Population)

- [1] Baseline is defined as the value obtained at the baseline visit.
- [2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC Sham, 6.0 x 10<sup>6</sup> hRPC Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix. This model incorporates missing data using multiple imputation

Programmer Note: Table 14.2.4.3.3 Mean Change in Contrast Sensitivity: Study Eye (EE Population)

- [1] Baseline is defined as the value obtained at the baseline visit.
- [2] Estimates of LS mean, LS mean difference (3.0 x 106 hRPC Sham, 6.0 x 106 hRPC Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix.

Table 14.2.5.1.1

Mean Change in Low Vision Functional Questionnaire (LV VA VFQ-48): Person mITT Population

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| Visual Ability at Baseline <sup>[1]</sup> | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | xx.x | XX X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Visual Ability at Month 6 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Change from Baseline to Month 6 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | XX, XX | xx, xx | XX, XX |
| LS Mean (SE) <sup>[2]</sup> | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| LS Mean Difference [95%CI] (SE) [2] | | xx x [xx x, xx.x] | xx x [xx x, xx x] |
| Visual Ability at Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x (xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| Change from Baseline to Month 12 | | | |
| n | n | n | n |
| Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx x (xx x) |
| Median | XX X | XX.X | XX X |
| Min, Max | xx, xx | xx, xx | XX, XX |
| LS Mean (SE) <sup>[2]</sup> | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| LS Mean Difference [95%CI] (SE) [2] | | xx x [xx x, xx.x] | xx x [xx x, xx x] |
| P-value <sup>[2]</sup> | | X.XXXX | X XXXX |

<sup>[1]</sup> Baseline is defined as the value obtained at the baseline visit.

[2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC – Sham, 6.0 x 10<sup>6</sup> hRPC – Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix.

path/t program.sas date time

Programmer Note: Continue table for Reading, Mobility, Visual information, Visual Motor for Visits: Month 6, Month 12.

Programmer Note: Table 14.2.5.1.2 Mean Change in Low Vision Functional Questionnaire: Study Eye using Multiple Imputation (mITT Population)

- [1] Baseline is defined as the value obtained at the baseline visit.
- [2] Estimates of LS mean, LS mean difference (3.0 x 10<sup>6</sup> hRPC Sham, 6.0 x 10<sup>6</sup> hRPC Sham), and two-sided p-values are obtained from a linear model for repeated measure. The model includes with visit, treatment, visit-by-treatment interaction and baseline as covariates, and unstructured covariance matrix. This model incorporates missing data using multiple imputation

Table 14.3.1 Study Drug Administration Safety Population

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| Eye Drug Injected into: | | | |
| OD (Right) | n (%) | n (%) | n (%) |
| OS (Left) | n (%) | n (%) | n (%) |
| Total Dose Administered | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Any Dose Interruptions | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Were any Adverse Events Observed? | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Subject Vital Signs Comparable to Pre Injection Levels | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Subject IOP < 30mm Post Treatment of Injection | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Subject Prescribed Topical Treatment after Study Drug | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |

path\t\_program.sas date time

Table 14.3.1.1
TEAEs by System Organ Class and Preferred Term
Safety Population

| System Organ Class / | Sham<br>(N=) | | | ) <sup>6</sup> hRPC<br>I=) | $6.0 \times 10^6 \text{ hRPC}$<br>(N=) | |
|---|---|---|---|---|---|---|
| Preferred Term | Subjects | Events | Subjects | Events | Subjects | Events |
| Subjects Reporting at Least One TEAE | n (%) | XX | n (%) | XX | n (%) | xx |
| System Organ Class 1 | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX |
| System Organ Class 2 | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX |

• • •

Programmer Note:sort table by Alphabetical SOC order, with in the SOC Alphabetical PT.

Table 14.3.1.2
TEAEs by System Organ Class, Preferred Term and Maximum Severity
Safety Population

| | Sham<br>(N=) | | | | $3.0 \times 10^6 \text{ hRPC}$<br>(N=) | | | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class / Preferred Term | Mild | Moderate | Severe | Life<br>Threatening | Death | Mild | Moderate | Severe | Life<br>Threatening | Death | Mild | Moderate | Severe | Life<br>Threatening | Death |
| Subjects Reporting at Least One TEAE | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) | n (%)<br>n (%)<br>n (%) |

<sup>.</sup> Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using maximum severity grade. path\t program.sas date time

Programmer Note:sort table by Alphabetical SOC order, with in the SOC Alphabetical PT.

jCyte, Inc.
Protocol: JC-02

Table 14.3.1.3
Related to Study Drug TEAEs by System Organ Class and Preferred Term
Safety Population

| System Organ Class / Preferred Term | Sha<br>(N | | $3.0 \times 10^6 \text{ hRPC}$<br>(N=) | | $6.0 \times 10^6 \text{ hRPC}$<br>(N=) | |
|---|---|---|---|---|---|---|
| | Subjects | Events | Subjects | Events | Subjects | Events |
| Subjects Reporting at Least One Related TEAE | n (%) | XX | n (%) | xx | n (%) | XX |
| System Organ Class 1 | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX |
| <br>System Organ Class 2 | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX |

.Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one adverse event are counted only once using the closest relationship to study drug.

Note: Related lincludes all events reported as "Possibly Related", "Related" or have missing relationship to study drug.

path\t program.sas date time

Programmer Note: sort table by Alphabetical SOC order, with in the SOC Alphabetical PT.

jCyte, Inc.
Protocol: JC-02

Table 14.3.1.4 Serious TEAEs by System Organ Class and Preferred Term Safety Population

| System Organ Class /<br>Preferred Term | Sha<br>(N= | $3.0 \times 10^{6} \text{ hRPC}$ (N=) | | $6.0 \times 10^6 \text{ hRPC}$<br>(N=) | | |
|---|---|---|---|---|---|---|
| | Subjects | Events | Subjects | Events | Subjects | Events |
| Subjects Reporting at Least One Serious TEAE | n (%) | xx | n (%) | xx | n (%) | xx |
| System Organ Class 1 | n (%) | XX | n (%) | xx | n (%) | xx |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX |
| System Organ Class 2 | n (%) | xx | n (%) | XX | n (%) | xx |
| Preferred Term 1 | n (%) | XX | n (%) | XX | n (%) | XX |
| Preferred Term 2 | n (%) | XX | n (%) | XX | n (%) | XX |

Note: At each level of summation (overall, system organ class, preferred term), subjects reporting more than one serious adverse event are counted only once. path\t\_program.sas date time

Programmer Note: sort table by Alphabetical SOC order, with in the SOC Alphabetical PT.

ocol: JC-02
Table 14.3.4.1
Hematology
Safety Population

| Laboratory Parameter | Time Point | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|---|
| Hemoglobin (g/dL), | Baseline [1] | | | |
| | n | n | n | n |
| | Mean (SD) | xx x (xx x) | xx x (xx x) | xx x (xx x) |
| | Median | xx x | xx x | XX X |
| | Min, Max | XX, XX | xx, xx | xx, xx |
| | Day 28 | | | |
| | N | n | n | n |
| | Mean (SD) | xx x (xx x) | xx x (xx x) | xx x (xx x) |
| | Median | xx x | xx x | XX X |
| | Min, Max | XX, XX | xx, xx | xx, xx |
| | Day 28 Change from Baseline | | | |
| | Ň | n | n | n |
| | Mean (SD) | xx x (xx x) | xx x (xx x) | xx x (xx x) |
| | Median | xx x | xx x | XX X |
| | Min, Max | xx, xx | XX, XX | xx, xx |
| | Month 3 | | | |
| | n | n | n | n |
| | Mean (SD) | xx x (xx x) | xx x (xx x) | xx x (xx x) |
| | Median | xx x | xx x | xx x |
| | Min, Max | XX, XX | XX, XX | XX, XX |

<sup>[1]</sup> Baseline is defined as the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date time

Programmer Note: Continue table for Visits: Day 28, Month 3, Month 6, Month 12/Early Termination.

Programmer Note: Table will include the following hematology parameters: Hemoglobin (g/dL), Hematocrit (%), Platelet Count(x  $10^9/L$ ), Red cell Count (x  $10^12/L$ ), White cell Count(x  $10^9/L$ ), Percent Neutrophil(%)s, Percent Lymphocytes(%)s, Percent Monocytes(x  $10^9/L$ ), Eosinophils(x  $10^9/L$ ), Monocytes (x  $10^9/L$ ). and Basophils(x  $10^9/L$ ).

Table 14.3.4.2 Chemistry Safety Population

| Laboratory Parameter | Time Point | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|---|
| ALT (SGPT) (U/L) | Baseline [1] | | | |
| | n | n | n | n |
| | Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx.x (xx.x) |
| | Median | xx x | xx.x | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| | Day 28 | | | |
| | Ň | n | n | n |
| | Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx.x (xx.x) |
| | Median | xx x | xx.x | XX.X |
| | Min, Max | xx, xx | XX, XX | xx, xx |
| | Day 28 Change from Baseline | | | |
| | N | n | n | n |
| | Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx.x (xx.x) |
| | Median | xx x | XX.X | xx.x |
| | Min, Max | xx, xx | XX, XX | xx, xx |
| | Month 3 | | | |
| | n | n | n | n |
| | Mean (SD) | xx x (xx x) | xx.x(xx.x) | xx.x (xx.x) |
| | Median | xx x | xx.x | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> Baseline is defined as the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date time

Programmer Note: Continue table for Visits: Day 28, Month 3, Month 6, Month 12/Early Termination.

Programmer Note: Table will include the following chemistry parameters: ALT (SGPT) (U/L), AST (SGOT) (U/L), Alkaline Phosphatase (U/L), Bilirubin (mg/dL), Sodium (mmol/L), Chloride (mmol/L), Carbon Dioxide (mmol/L), Blood Urea Nitrogen (mg/dL), Creatinine (mg/dL), Total Protein (g/dL), Albumin (g/dL), Calcium(mg/dL), Phosphate (mg/dL), Glucose (mg/dL) and HbA1c (%).

Table 14.3.4.3 Vital Signs Safety Population

| Vital Sign | Time Point | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|---|
| Systolic BP (mmHg) | Day 0 15 min Post-Injection (Baseline) [1] | | | |
| | n | n | n | n |
| | Mean (SD) | xx x (xx x) | xx x (xx x) | xx.x (xx.x) |
| | Median | XX X | XX X | xx.x |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | Day 0 15 min Post-Injection | | | |
| | n | n | n | n |
| | Mean (SD) | xx x (xx x) | xx x (xx x) | xx.x (xx.x) |
| | Median | XX X | XX X | xx.x |
| | Min, Max | XX, XX | XX, XX | XX, XX |

<sup>[1]</sup> Baseline is defined as the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date time

Programmer Note: Table will include the following vital signs: systolic BP (mmHg), diastolic BP (mmHg), Heart Rate (bpm), Respiration (Breaths/min) and Temperature(°C).

Programmer Note: Continue table for Visits: Day0-15min Post-Injection, Day 0-60 min post injection, Day 1, Day 28, Month 3, Month 6, Month 9, Month 12/Early Termination.

Table 14.3.4.4.1 Slit Lamp Examination: Study Eye Safety Population

| | Sham | $3.0 \times 10^6 \mathrm{hRPC}$ | 6.0 x 10 <sup>6</sup> hRPC |
|---|---|---|---|
| | (N=) | (N=) | (N=) |
| Eyelids | | | |
| Baseline [1] | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |
| Day 1 | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |
| Day 7 | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |
| Day 28 | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |
| Month 3 | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |

<sup>[1]</sup> Baseline is defined as the last non-missing value recorded prior to the first dose of study drug.

path\t\_program.sas date time

Programmer Note: Continue table for Eyelashes, Conjunctiva, Sclera, Cornea, Anterior Chamber Flare), Iris, Lens Status, Cataract Type, Grade.

Programmer Note: Continue table for Visits: Day 1, Day 7, Day 28, Month 3, Month 6, Month 9, Month 12.

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that Particular time point...

Programmer Note: Table can be modified to align with information collected on the CRF.

<sup>[2]</sup> Subject may be counted more than one row.

**Table 14.3.4.4.1** Slit Lamp Examination: Study Eye **Safety Population** 

| | Sham | $3.0 \times 10^6 hRPC$ | $6.0 \times 10^{6} \text{ hRPC}$ |
|---|---|---|---|
| | (N=) | (N=) | (N=) |
| Lens Status | | | |
| Baseline [1] | (n=) | (n=) | (n=) |
| Aphakic | n (%) | n (%) | n (%) |
| Psedophakic | n (%) | n (%) | n (%) |
| Phakic | n (%) | n (%) | n (%) |
| Day 1 | (n=) | (n=) | (n=) |
| Aphakic | n (%) | n (%) | n (%) |
| Psedophakic | n (%) | n (%) | n (%) |
| Phakic | n (%) | n (%) | n (%) |
| Cataract Type [2] | | | |
| Baseline [1] | (n=) | (n=) | (n=) |
| Nuclear | n (%) | n (%) | n (%) |
| Cortical | n (%) | n (%) | n (%) |
| Posterior Subcapsular | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) |
| Day 1 | (n=) | (n=) | (n=) |
| Nuclear | n (%) | n (%) | n (%) |
| Cortical | n (%) | n (%) | n (%) |
| Posterior Subcapsular | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) |
| Grade | | | |
| Baseline [2] | (n=) | (n=) | (n=) |
| +1 | n (%) | n (%) | n (%) |
| +2 | n (%) | n (%) | n (%) |
| +3 | n (%) | n (%) | n (%) |
| +4 | n (%) | n (%) | n (%) |

<sup>[1]</sup> Baseline is defined as the last non-missing value recorded prior to the first dose of study drug.

path\t\_program.sas date time

Programmer Note: Continue table for Eyelashes, Conjunctiva, Sclera, Cornea, Anterior Chamber Flare), Iris, Lens Status, Cataract Type, Grade.. Programmer Note: Continue table for Visits: Day 1, Day 7, Day 28, Month 3, Month 6, Month 9, Month 12.

<sup>[2]</sup> Subject may be counted more than one row.

Programmer Note: Table 14.3.4.4.2 will contain the same information for the Non-Study Eye.

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that particular time point.

Programmer Note: Table can be modified to align with information collected on the CRF.

Table 14.3.4.5.1 Intraocular Pressure (IOP): Study Eye **Safety Population** 

| | Sham<br>(N=) | $3.0 \times 10^6 \text{ hRPC}$<br>(N=) | $6.0 \times 10^6 \text{ hRPC}$<br>(N=) |
|---|---|---|---|
| - | ( ) | () | (- ) |
| Baseline [1] | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx x (xx x) | xx x (xx x) |
| Median | xx.x | XX X | XX X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| Day 0 | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx x (xx x) | xx x (xx x) |
| Median | XX.X | XX X | XX X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| Day 0 Change from Baseline | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx x (xx x) | xx x (xx x) |
| Median | XX.X | XX X | XX X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| Day 1 | | | |
| n | n | n | n |
| Mean (SD) | xx.x (xx.x) | xx x (xx x) | xx x (xx x) |
| Median | xx.x | xx x | xx x |
| Min, Max | xx, xx | xx, xx | xx, xx |

<sup>[1]</sup> Baseline is defined as the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date time

Programmer Note: Continue table for Visits: Day 1, Day 7, Day 28, Month 3, Month 6, Month 9, Month 12. Programmer Note: Table 14.3.4.5.2 will contain the same information for the Non-Study Eye.

> **Table 14.3.4.6.1 B-Scan: Study Eye Safety Population**

| | Sham<br>(N=) | $3.0 \times 10^6 \text{ hRPC}$<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| - | | | ( ) |
| Baseline [1] | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |
| Good | n (%) | n (%) | n (%) |
| Poor | n (%) | n (%) | n (%) |
| Injected Cells Visualized | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Not Applicable | n (%) | n (%) | n (%) |
| Day 7 | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |
| Good | n (%) | n (%) | n (%) |
| Poor | n (%) | n (%) | n (%) |
| Injected Cells Visualized | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Not Applicable | n (%) | n (%) | n (%) |

<sup>[1]</sup> Baseline is defined as the last non-missing value recorded prior to the first dose of study drug. path\t program.sas date

Programmer Note: Continue table for Visits: Day 7, Month 6 and Month 12.

Programmer Note: Table 14.3.4.6.2 will contain the same information for the Non-Study Eye

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that particular time point.

Table 14.3.4.7.1
Dilated Fundoscopic Examination :Study Eye
Safety Population

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| Vitreous Examination | | | |
| Baseline [1] | (n=) | (n=) | (n=) |
| Mild +1 | n (%) | n (%) | n (%) |
| Moderate +2 | n (%) | n (%) | n (%) |
| Severe +3 | n (%) | n (%) | n (%) |
| Very Severe +4 | | | |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |
| Day 1 | (n=) | (n=) | (n=) |
| Mild +1 | n (%) | n (%) | n (%) |
| Moderate +2 | n (%) | n (%) | n (%) |
| Severe +3 | n (%) | n (%) | n (%) |
| Very Severe +4 | | | |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |
| Day 7 | (n=) | (n=) | (n=) |
| Mild +1 | n (%) | n (%) | n (%) |
| Moderate +2 | n (%) | n (%) | n (%) |
| Severe +3 | n (%) | n (%) | n (%) |
| Very Severe +4 | | | |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |

<sup>[1]</sup> Baseline is defined as the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date time

Programmer Note: Continue table for Optic Nerve, Macula, and Peripheral Retina Examinations. Programmer Note: Continue table for Visits:, Day 7, Day 28, Month 3, Month 6, Month 9, Month 12.

Programmer Note: Table 14.3.4.7.2 will contain the same information for the Non-Study Eye.

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point.

**Table 14.3.4.8** Post Injection Clinical Vitreous Exam: Study Eye **Safety Population** 

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | $6.0 \times 10^6 \text{ hRPC}$<br>(N=) |
|---|---|---|---|
| | (11) | (14-) | (11-) |
| Day0 | (n=) | (n=) | (n=) |
| Injected eye examined | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Methods of Examination [1] | | | |
| Indirect Ophthalmoscopy | n (%) | n (%) | n (%) |
| Fundus Exam | n (%) | n (%) | n (%) |
| Slit Lamp Exam | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) |
| Change from Previous Exam | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |
| Appearance | | | |
| Cells | n (%) | n (%) | n (%) |
| Clumps | n (%) | n (%) | n (%) |
| Opacity | n (%) | n (%) | n (%) |
| Debris | n (%) | n (%) | n (%) |
| Strands | n (%) | n (%) | n (%) |
| Inflammation | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) |
| Photograph taken | | | |
| Yes | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) |

<sup>[1]</sup> Subject may be counted more than one row.

path\t program.sas date time .

Programmer Note: Continue table for Visits: Day 1, Day 7, Day 28, Month 3, Month 6, Month 9, and Month 12.

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that particular time point.

Table 14.3.4.9.1 Optical Coherence Tomography (OCT): Study Eye Categorical Analysis
Safety Population

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| Cystoid Macular Edema (CME) present | | | |
| Baseline [1] | n/N (%) | n/N (%) | n/N (%) |
| Month 6 | n/N (%) | n/N (%) | n/N (%) |
| Month 12 | n/N (%) | n/N (%) | n/N (%) |
| If CME Present, Involve Foveal Center | | | |
| Baseline [1] | n/N (%) | n/N (%) | n/N (%) |
| Month 6 | n/N (%) | n/N (%) | n/N (%) |
| Month 12 | n/N (%) | n/N (%) | n/N (%) |
| Epiretinal Membrane Formation Present | | | |
| Baseline [1] | n/N (%) | n/N (%) | n/N (%) |
| Month 6 | n/N (%) | n/N (%) | n/N (%) |
| Month 12 | n/N (%) | n/N (%) | n/N (%) |
| Evidence of Retinal Traction | | | |
| Baseline [1] | n/N (%) | n/N (%) | n/N (%) |
| Month 6 | n/N (%) | n/N (%) | n/N (%) |
| Month 12 | n/N (%) | n/N (%) | n/N (%) |

<sup>[1]</sup> Baseline is defined as the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date

Programmer Note: Continue table for Visits: Month 6, Month 12..

Programmer Note: Table 14.3.4.9.2 will contain the same information for the Non-Study Eye

Table 14.3.4.10.1 Autofluorescence : Study Eye Safety Population

| | Sham<br>(N=) | 3.0 x 10 <sup>6</sup> hRPC<br>(N=) | 6.0 x 10 <sup>6</sup> hRPC<br>(N=) |
|---|---|---|---|
| Baseline [1] | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |
| Month 6 | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |
| Month 12 | (n=) | (n=) | (n=) |
| Normal | n (%) | n (%) | n (%) |
| Abnormal, Not Clinically Significant | n (%) | n (%) | n (%) |
| Abnormal, Clinically Significant | n (%) | n (%) | n (%) |

<sup>[1]</sup> Baseline is defined as the value obtained at the baseline visit. If the baseline value is missing, the baseline value will be the last non-missing value recorded prior to the first dose of study drug. path\t\_program.sas date time

Programmer Note: Continue table for Visits:.Month 6, Month 12.

Programmer Note: Denominators used for percentage calculation to be based on number of results reported for that perticular time point.

Programmer Note: Table 14.3.4.10.2 will contain the same information for the Non-Study Eye.
Appendix D: Listing Layouts

RUC Error! AutoText entry not defined.

### Listing 16.2.1.1 Subject Disposition All Subjects

Actual Subject Treatment Information Study Drug Completion or Primary Reason for Subject Randomized Subject Study Eye Safety ITT Consent Date Administration Discontinuation Population [1] Population [2] Treatment Group ID Received Date/Time Date Discontinuation OD Sham Yes Yes/No Yes/No IS08601 ISO8601 IS08601 xxx--xxx xxxxxxxxxxxxxxx (Right) .  $3.0 \times 10^6 \text{ hRPC}$ Yes OS (Left) Yes/No Yes/No ISO8601 ISO8601 ISO8601 XXX--XXX XXXXXXXXXXXXXXXX .  $6.0 \times 10^6 \text{ hRPC}$  xxx--xxx ISO8601 Yes OS (Left) Yes/No Yes/No ISO8601 ISO8601 XXXXXXXXXXXXXXXX

Note: Randomization Treatment displayed in Treatment Group column.

path\l program.sas date time

Programmer Note: Include Reasons, Death and AE # information in "Primary Reason for Discontinuation" column.

<sup>[1]</sup> Received any amount of study treatment (including sham).

<sup>[2]</sup> All randomized subjects who provide any post-randomization data.

jCyte, Inc.
Protocol: JC-02

### Listing 16.2.2.1 Protocol Deviations All Subjects

| Treatment<br>Group | Subject<br>ID | Deviation<br>Date | Date<br>Identified | Protocol<br>Deviation<br>Category | Description of Protocol Deviation | Significant<br>Deviations | Deviation<br>Detail |
|---|---|---|---|---|---|---|---|
| Sham | xxxxxx | ISO8601 | ISO8601 | xxxxxxxx | xxxxxxxx | xxxxx | xxxxx |
| 3.0 x 10 <sup>6</sup> hRP | C xxxxxx | | | xxxxxxxx | xxxxxxxx | | |
| .6.0 x 10 <sup>6</sup><br>hRPC | xxxxxx | | | xxxxxxxx | xxxxxxxx | | |

path\l\_program.sas date time

jCyte, Inc. Protocol: JC-02 Page 1 of x

## Listing 16.2.2.2 Inclusion/Exclusion Criteria All Subjects

| Treatment Group | Subject<br>ID | All Eligibility<br>Criteria Met? | If Not Met,<br>Inc/Exc Criterion ID Not Met |
|---|---|---|---|
| Sham | xxxxxx | Yes/No | Inclusion #/Exclusion# |
| 3.0 x 10 <sup>6</sup> hRPC | xxxxxx | Yes/No | Inclusion #/Exclusion# |
| 6.0 x 10 <sup>6</sup> hRPC | xxxxxx | Yes/No | Inclusion #/Exclusion# |

path\l\_program.sas date

Listing 16.2.4.1
Demographic and Baseline Characteristics **Safety Population** 

| Treatment Group | Subject ID | Date of<br>Birth | Age<br>(years) | Sex | If Female,<br>Childbearing<br>Potential? | If YES,<br>Method of<br>Birth Control | If No, Why is<br>Subject not of<br>Childbearing<br>Potential? | Ethnicity | Race | Baseline<br>Height<br>(cm) | Baseline<br>Weight<br>(Kg) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Sham | xxxxxx | ISO8601 | xx | Female | No/Yes | IUD | Surgical<br>Sterilization | Hispanic<br>or Latino | Asian | xxx | xxx |
| | xxxxxx | ISO8601 | XX | Male | No/Yes | Oral<br>Contraception | Post Menopausal | Not<br>Hispanic<br>or Latino | White | xxx | xxx |
| | <br>xxxxxx | ISO8601 | xx | Female | No/Yes | Other: Specify | Other: Specify | Hispanic<br>or Latino | Black or<br>African<br>American | xxx | XXX |

path\l\_program.sas date time

Programmer Note: Include Specification for Other in "Method of Birth Control" column if applicable

**Listing 16.2.4.2** Medical History Safety Population

| Treatment Group | Subject ID | MH# | Body System | Medical History Condition/Event | Start Date | End Date/Ongoing |
|---|---|---|---|---|---|---|
| Sham | xxxxxx | 1 | xxxxxxx | xxxxxxxxxx | ISO8601 | ISO8601./Ongoing |
| $3.0 \times 10^6 \text{hRPC}$ | xxxxxx | 2 | xxxxxxx | xxxxxxxxxxx | ISO8601 | ISO8601./Ongoing |
| $6.0 \times 10^6 \text{hRPC}$ | xxxxxx | 2 | xxxxxxxx | xxxxxxxxxxx | ISO8601 | ISO8601./Ongoing |

path\l\_program.sas date time

Programmer Note: sort by medical history number within each subject.
Programmer Note: If MH marked as Ongoing, then show "Ongoing" under End Date column.

### Listing 16.2.4.3 Ocular Medical History Safety Population

| Treatment Group | Subject ID | Ocular<br>MH # | Eye | Body System | Ocular MH<br>Condition/Diagnosis/Surgery | Date of<br>Diagnosis/Surgery | Date Resolved/Ongoing |
|---|---|---|---|---|---|---|---|
| Sham | xxxxxx | 1 | OD | xxxxxxxxxxxx | xxxxxxxxxxx | ISO8601 | ISO8601./Ongoing |
| 3.0 x 10 <sup>6</sup> hRPC | xxxxxx | 1 | OS | xxxxxxxxxxx | xxxxxxxxxxx | ISO8601 | ISO8601./Ongoing |
| $6.0 \times 10^6 \text{hRPC}$ | xxxxxx | 1 | OS | xxxxxxxxxxxx | xxxxxxxxxxx | ISO8601 | ISO8601./Ongoing |

path\l\_program.sas date time

Programmer Note: sort by medical history number within each subject.

Programmer Note: If MH marked as ongoing end date, then show "Ongoing" under Date Resolved column...

Page 1 of x jCyte, Inc. Protocol: JC-02

Listing 16.2.5 Study Drug Administration Safety Population

| Treatment | Subject ID | | Date and Time | | Not Done: | | Dose<br>Interruptions? | AEs | Vital Signs<br>comparable to<br>Pre-Treatment of<br>Study drug | of Study Drug | Prescribed<br>Topical<br>Treatment after<br>Treatment of<br>Study Drug |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | (Study Eye) | Visit | of Injection | Time | Reason | ? Reason | Reason | Observed? | Injection | Injection | Injection |
| Sham | Xxxxx (OS) | Day 0 | ISO8601 | ISO8601 | | Yes | Yes: Reason | No/Yes | No/Yes | No/Yes | No/Yes |
| 3.0 x 10 <sup>6</sup> hRPC | Xxxxx (OS) | Day 0 | ISO8601 | | | No: Reason | Yes: Reason | No/Yes | No/Yes | No/Yes | No/Yes |
| 6.0 x 10 <sup>6</sup> hRPC | Xxxxx (OS) | Day 0 | ISO8601 | | | Yes | Yes: Reason | No/Yes | No/Yes | No/Yes | No/Yes |

path\l\_program.sas date time

Listing 16.2.6.1
Best Corrected Visual Acuity (ETDRS and/or FrACT)
ITT Population

| | | | | | | | OD Visual Acu | ıity | OS V | Visual Acu | ity |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatmen<br>t Group | Subje<br>t<br>ID | c<br>Visit | Assessme<br>nt<br>Date | Study<br>Day | Not Done:<br>Reason | Measurem<br>ent | BCVA<br>Method Used | Total<br>Numbers of<br>Letters<br>Correct | Measurement | BCVA<br>Method<br>Used | Total<br>Numbers of<br>Letters<br>Correct |
| Sham | XXX-<br>XXX | ng | ISO8601 | xx | | Xx/xxx | E-ETDRS | xxx | Xx/xxx | E-<br>ETDRS | xxx |
| | | Baselin<br>e | | | | Xx/xxx | | XXX | Xx/xxx | | XXX |
| | | Day0 | | | | Xx/xxx | | XXX | Xx/xxx | | XXX |
| | | Day1 | | | | Xx/xxx | | XXX | Xx/xxx | | XXX |
| | | Day7 | | | | Xx/xxx | | XXX | Xx/xxx | | XXX |
| | | Day28 | | | | Xx/xxx | | XXX | Xx/xxx | | XXX |
| | | Month3 | 1 | | | Xx/xxx | | XXX | Xx/xxx | | XXX |
| | | Month6 | • | | | $X_{X}/x_{X}$ | | XXX | Xx/xxx | | XXX |
| | | Month9 | | | | Xx/xxx | | XXX | Xx/xxx | | XXX |
| | | Month 1<br>2/Early<br>Termin<br>ation | | | | Xx/xxx | | XXX | Xx/xxx | | XXX |
| 3.0 x 10 <sup>6</sup><br>hRPC | XXX-<br>XXX | Screeni<br>ng, | | | | | FrACT | | | FrACT | |
| 6.0 x 10 <sup>6</sup><br>hRPC | XXX-<br>XXX | Screeni<br>ng, | | | | | FrACT | | | FrACT | |

path\l\_program.sas date

time

Listing 16.2.6.2 Optical Coherence Tomography (OCT) Safety Population

| | | | | Study Day | Not Done: Reason | | | Was There | If Yes, Was There |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Cystoid Macular | IF CME Present, | Epiretinal | Evidence of Retinal |
| | | | Assessment | | | Edema (CME) | Involve Foveal | Membrane | Traction? |
| Treatment Group | Subject ID | Visit | Date | | | Present? | Center? | Formation Present? | |
| Sham | xxxxxx | Baseline | ISO8601 | XX | | Yes/No | Yes/No | Yes/No | Yes/No |
| | | Month 6 | ISO8601 | XX | | Yes/No | Yes/No | Yes/No | Yes/No |
| | | Month 12/Early<br>Termination | ISO8601 | XX | | Yes/No | Yes/No | Yes/No | Yes/No |
| 3.0 x 10 <sup>6</sup> hRPC | xxxxxx | Baseline | | XX | | Yes/No | Yes/No | Yes/No | Yes/No |
| 5.0 H 10 HH 0 | | Month 6 | | XX | | Yes/No | Yes/No | Yes/No | Yes/No |
| | | Month 12/Early<br>Termination | | XX | | Yes/No | Yes/No | Yes/No | Yes/No |
| 6.0 x 10 <sup>6</sup> hRPC | xxxxxx | Baseline | | XX | | Yes/No | Yes/No | Yes/No | Yes/No |
| mu | | Month 6 | | XX | | Yes/No | Yes/No | Yes/No | Yes/No |
| | | Month 12/Early | | XX | | Yes/No | Yes/No | Yes/No | Yes/No |
| | | Termination | | | | | | | |

path\l\_program.sas date time

Listing 16.2.6.3 Autofluorescence Safety Population

| Treatment Group | Subject ID | Visit | Assessment<br>Date | Study Day | Not Done: Reason | Right Eye (OD)<br>Result | Left Eye (OS) Result |
|---|---|---|---|---|---|---|---|
| C1 | | D 1' | 1000601 | | | N. 1 | N. 1 |
| Sham | XXXXXX | Baseline | ISO8601 | XX | | Normal | Normal |
| | | Month 6 | ISO8601 | XX | | Abnormal CS: Abnormality | Abnormal CS:Abnoramlity |
| | | Month 12/Early<br>Termination | ISO8601 | XX | | Abnormal NCS: | Abnormal NCS |
| 3.0 x 10 <sup>6</sup> hRPC | xxxxxx | Baseline | ISO8601 | XX | | Normal | Normal |
| | | Month 6 | ISO8601 | XX | | Abnormal CS<br>Abnormality | Abnormal CS: Abnormality |
| | | Month 12/Early<br>Termination | ISO8601 | xx | | Abnormal NCS | Abnormal NCS |
| 6.0 x 10 <sup>6</sup> hRPC | xxxxxx | Baseline | ISO8601 | XX | | Normal | Normal |
| | | Month 6 | ISO8601 | XX | | Abnormal CS<br>Abnormality | Abnormal CS: Abnormality |
| | | Month 12/Early<br>Termination | ISO8601 | XX | | Abnormal NCS | Abnormal NCS |

Note: CS=Clinically Significant, NCS=Not Clinically Significant.

path\l\_program.sas date time

Programmer Note: Include Description of Abnormality and Clinically Significant information in "Result" column

Listing 16.2.6.4 Visual Field ITT Population

| | | | | | | | OD (Right) | | | | | | OS (L | eft) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatm | | | Assessmer | n<br>Study | | Not | Reactio | Stimulus Island a | # | Visual<br>Field | | | Reaction<br>Time<br>(ms) | | | Visual<br>Field<br>Area or | |
| ent<br>Group | Subject | Visit | Date and<br>Time | • | End<br>Time | Done: | Fixation n Time<br>Stability (ms) | Size | | Area or<br>Island | Sum | Fixation<br>Stability | . , | Stimulus<br>Size | Island Quadran<br># t | | Sum |
| Sham | xxxxxx | Baseline | ISO8601 | xx | ISO86<br>01 | | 1 | III4e | A | xxx.x | | 1 | | III4e | A | xxx x | |
| | | Month 6 | ISO8601 | XX | | | 2 | I4e | В | XXX.X | | 2 | No | I4e | В | XXX X | |
| | | Month 12 | | XX | | | 3 | V4e | C | xxx.x | | 3 | | V4e | C | xxx x | |
| 3.0 x<br>10 <sup>6</sup><br>hRPC | xxxxxx | Baseline | | xx | | | 4 | Other | D | XXX.X | | 4 | | III4e | D | xxx x | |
| iiki C | | Month 6 | | | | | 5 | I4e | Е | XXX.X | | 5 | | I4e | E | xxx x | |
| | | Month 12 | | | | | 1 | V4e | A | XXX.X | | 1 | Not | V4e | A | XXX X | |
| | | Wionui 12 | 2 | | | | ı | V 4C | A | AAA.A | | 1 | Applicabl<br>e | | A | AAA A | |
| 6.0 x<br>10 <sup>6</sup><br>hRPC | xxxxxx | Baseline | | | | | 4 | Other | D | XXX.X | | 4 | | III4e | D | xxx x | |
| IIKPC | | Month 6 | | | | | 5 | I4e | Е | XXX.X | | 5 | | I4e | Е | xxx x | |
| | | Month 12 | | | | | 1 | V4e | A | XXX.X | | 1 | Not | V4e | Ā | XXX X | |
| | | | _ | | | | - | | | | | - | Applicabl e | | | | |

Note: A=Central, B=Upper Right, C=Lower Right, D=Lower Left, E=Upper Left.

Note: 1=Unable to find fixation target, 2=Able to maintain fixation 25% of the time, 3=Able to maintain fixation 50% of the time, 4=Able to maintain fixation 75% of the time, 5=Able to maintain fixation 100% of the time.

path\l\_program.sas date time

Programmer Note: there will be multiple islands at each timepoint. Programmer Note: Visual Field area is same as Adjusted calculated Sized in CRF.

Programmer Note: Sum will be calculated using for a subject with same visit, same date and time with same stimulus size then sum all the adjusted calculate size and put the value in first row of that visit.

jCyte, Inc. Protocol: JC-02 Page 1 of x

Listing 16.2.6.5 Mobility ITT Population

| Treatment<br>Group | Subject<br>ID | Visit | Assess<br>ment<br>Date | Study<br>Day | Not<br>Done:<br>Reason | Dark<br>Adapt | Dark<br>Adaption<br>Start Time | Dark<br>Adaption<br>End Time | Eye | Maximum<br>Step Speed | Illumination<br>Level | Converted<br>Scale<br>Score | Was Assessment<br>Done in more than<br>one Eye? | Eye | Maximum<br>Step Speed | | Converted<br>Scale<br>Score |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sham | xxxxxx | Baseline | eISO860 | xx | | Yes/No | ISO8601 | ISO8601 | Right<br>(OD) | XX | XX | | Yes/No | Right<br>(OD) | XX | XX | |
| | | Month 6 | 5 | XX | | | | | . , | XX | XX | | | ` ' | XX | XX | |
| | | Month<br>12 | ISO860<br>1 | XX | | | | | | XX | XX | | | | XX | XX | |
| 3.0 x 10 <sup>6</sup><br>hRPC | xxxxxx | Baseline | eISO860 | xx | | | | | Left (OS) | xx | XX | | Yes/No | Left (OS) | XX | XX | |
| | | Month 6 | 5 | XX | | | | | | XX | XX | | | | XX | XX | |
| | | Month<br>12 | | XX | | | | | | XX | XX | | | | XX | XX | |
| $6.0 \times 10^6$<br>hRPC | xxxxxx | Baseline | e | xx | | | | | Right<br>(OD) | XX | XX | | Yes/No | Right<br>(OD) | XX | XX | |
| | | Month 6 | 5 | XX | | | | | | XX | XX | | | | XX | XX | |
| | | Month<br>12 | | XX | | | | | | XX | XX | | | | XX | XX | |

path\l\_program.sas date time

### Listing 16.2.6.6 Contrast Sensitivity (CS) ITT Population

OD (Right)

| | | | | | | | | | ( | 0) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | | OS (Left) | |
| | | | | Study Day | Not | | | | Threshold | | | | | Threshol | |
| | | | | | Done: | | | | CS Value | Threshol | | | | d CS Thresho | |
| | | | Assessmen | t | Reason | | | | Number | d Value | Mean | | | Value ld Value | Mean |
| Treatment | | | Date and | | | | Spatial | | | | | Spatial | | Number | |
| Group | Subject ID | ) Visit | Time | | | End Time | Frequency | CS | | | | Frequency | CS | | |
| Sham | XXXXXX | Baseline | ISO8601 | XX | | ISO8601 | 1 | | | | | 1 | | | |
| | | Month 6 | ISO8601 | XX | | ISO8601 | 2 | | | | | 2 | | | |
| | | Month 12 | ISO8601 | XX | | | 3 | | | | | 3 | | | |
| $3.0 \times 10^6$ | XXXXXX | Baseline | ISO8601 | XX | | ISO8601 | 1 | | | | | 1 | | | |
| hRPC | | | | | | | _ | | | | | | | | |
| | | | | XX | | ISO8601 | 2 | | | | | 2 | | | |
| | | Month 12 | ISO8601 | XX | | | 3 | | | | | 3 | | | |
| 6.0 1.06 | | D 11 | 1000601 | | | 1000601 | | | | | | 4 | | | |
| $6.0 \times 10^6$ | XXXXXX | Baseline | ISO8601 | | | ISO8601 | 4 | | | | | 4 | | | |
| hRPC | | Month 6 | 1000601 | | | ISO8601 | 5 | | | | | 5 | | | |
| | | Month 6 | | | | | 5 | | | | | 3<br>1 | | | |
| | | Month 12 | 1209001 | | | ISO8601 | 1 | | | | | 1 | | | |

Note: If no value in threshold cs value, no mean is calculated. path\l\_program.sas date time

Programmer Note: for Threshold values, take first OECS3 value and next rows with OETHRVAL.

Programmer Note: for mean calculations, take first OECS3 value and add it to all OETHRVAL and take mean of those all values. If only one value in OECS3 and no values in OETHRVAL, then ignore that value and do not include in calculating mean.

Listing 16.2.6.7 Low Vision Functional Questionnaire (LV VA-VFQ-48) ITT Population

| | Subject | | Assessment<br>Date and | Study<br>Day | | Not Done:<br>Reason | Visual | | | Visual | Visual | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | - | isit | Time | Day | End Time | Keason | Ability | Reading | Mobility | Information | Motor | Comments |
| Sham | xxxxxx Basel | ine | ISO8601 | XX | ISO8601 | | XXX | XXX | XXX | XXX | XXX | XXX |
| | Mont | h 6 | ISO8601 | XX | | | XXX | XXX | XXX | XXX | XXX | XXX |
| | Mont | h 12 | ISO8601 | XX | | | XXX | XXX | XXX | XXX | XXX | XXX |
| $3.0 \times 10^6 hRPC$ | xxxxxx Basel | ine | ISO8601 | xx | | | xxx | xxx | xxx | XXX | xxx | XXX |
| | Mont | h 6 | | XX | | | XXX | XXX | XXX | XXX | XXX | XXX |
| | Mont | h 12 | | XX | | | XXX | XXX | XXX | XXX | XXX | XXX |
| $6.0 \times 10^6 \text{hRPC}$ | xxxxxx Basel | ine | | XX | | | xxx | XXX | xxx | xxx | XXX | XXX |
| | Mont | h 6 | | XX | | | xxx | xxx | xxx | XXX | xxx | XXX |
| | Mont | h 12 | | XX | | | XXX | XXX | XXX | xxx | XXX | xxx |

path\l\_program.sas date time

Listing 16.2.7.1 Adverse Events Safety Population

| | | | | Saf | ety Population | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Verbatim Term | Onset Date | | | | | | | |
| | | // System Organ | and Time | | | | Relationship | | Dose | |
| | Subject | Class//Preferred | (Study | End Date | | | to Study | Treatment | Limiting | |
| Treatment Group | ID | AE# Term | Day) | (Study Day) | Serious | Severity | Drug | of Event | Toxicity | Outcome |
| Sham | xxxxxx | | ISO8601(x<br>x) | ISO8601 (xx) | Yes | Mild | Not Related | None | Yes/No | Recovery/Resolved |
| | | | ISO8601(x<br>x) | ISO8601(xx) | No | Moderate | Unlikely<br>Related | Medication | Yes/No | Recovery/Resolved<br>W/Seq |
| | | | ISO8601(x<br>x) | ISO8601(xx) | No | Moderate | Possibly<br>Related | Non-Drug<br>Treatment | Yes/No | Recovering/Resolvi<br>ng |
| | | | ISO8601(x<br>x) | ISO8601(xx) | No | Mild | Related | Hospitalization | Yes/No | Not<br>Recovered |
| | | | ISO8601(x x) | ISO8601 (xx) | No | Severe | Unlikely<br>Related | | Yes/No | Fatal |
| | | | ISo8601(x<br>x) | ISO8601(xx) | No | Mild | | | | |
| | | • | | | | | | | | |
| 3.0 x 10 <sup>6</sup> hRPC | xxxxxx | | | | | | | | | |

6.0 x 10<sup>6</sup> hRPC xxx--xxx

.....

path\l\_program.sas date time

Programmer Note: sort by subject and AE # subject

### Listing 16.2.7.2 Serious Adverse Events Safety Population

| Treatment Group | Subject<br>ID | Verbatim Term // System Organ AE Class//Preferred # Term | Onset Date<br>and Time<br>(Study Day) | End Date<br>(Study Day) | Severity | Relationship<br>to Study Drug | Treatment of Event | Dose Limiting<br>Toxicity | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| Sham | xxxxxx | | ISO8601<br>(xx) | ISO8601(xx) | Mild | Not Related | None | Yes/No | Recovery/Resolve |
| | | | ISO8601<br>(xx) | ISO8601 (xx) | Moderate | Unlikely<br>Related | Medication | Yes/No | Recovery/Resolve<br>d W/Seq |
| | | | ISO8601<br>(xx) | ISO8601 (xx) | Moderate | Possibly<br>Related | Non-Drug<br>Treatment | Yes/No | Recovering/Resol ving |
| | | | ISO8601<br>(xx) | ISO8601 (xx) | Mild | Related | Hospitalization | Yes/No | C |
| | | | ISO8601<br>(xx) | ISO8601 (xx) | Severe | Unlikely<br>Related | | | |
| | | | ISO8601<br>(xx) | ISO8601 (xx) | Mild | | | | |
| 3.0 x 10 <sup>6</sup> hRPC | xxxxxx | | | | | | | | |
| 6.0 v 106 hDDC | VVV VVV | | | | | | | | |

 $6.0 \times 10^6 \text{ hRPC}$   $\times \times \times -\times \times$ 

path\l\_program.sas date time

Programmer Note: sort by subject and AE # subject

**Listing 16.2.7.3** Related Adverse Events **Safety Population** 

| | | | | Onset | | | | | | Dose Limiting | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Subject | ΑE | Verbatim Term // System Organ | Date/Time | End Date | | | Relationship | Treatment | Toxicity | |
| Treatment Group | ID | # | Class// Preferred Term | (Study Day) | (Study Day) | Serious | Severity | to Study Drug | of Event | | Outcome |
| Sham | xxxxxx | 1 | Xxxxxxxxx//xxxxxxxx//xxxxxx | ISO8601.(xx) | ISO8601.(xx) | Yes | Mild | Related | None | Yes/No | Recovery/Resolved |
| Sildin | AAA AAA | 2 | Xxxxxxxxx//xxxxxxx//xxxxxx | ISO8601.(xx) | ISO8601.(xx) | No | Moderate | Related | Medication | Yes/No | Recovery/Resolved<br>W/Seq |
| | | 3 | Xxxxxxxxx//xxxxxxxx//xxxxxx | ISO8601.(xx) | ISO8601.(xx) | No | Moderate | Possibly Related | Non-Drug<br>Treatment | Yes/No | Recovering/Resolv ing |
| | | 4 | Xxxxxxxxx//xxxxxxxx//xxxxxx | ISP8601.(xx) | ISO8601.(xx) | No | Mild | Related | Hospitalizat ion | Yes/No | C |
| | | 5 | Xxxxxxxxx//xxxxxxxx//xxxxxx | ISO8601.(xx) | ISO8601.(xx) | Yes | Severe | Related | | | |
| | | 6 | Xxxxxxxxx//xxxxxxxx//xxxxxx | ISO8601.(xx) | ISO8601.(xx) | No | Mild | | | | |
| | | 7 | Xxxxxxxxxx//xxxxxxxx//xxxxxx | ` ´ | ` ´ | | | | | | |
| | | 8 | Xxxxxxxxxx//xxxxxxxx//xxxxxx | | | | | | | | |
| 3.0 x 10 <sup>6</sup> hRPC | xxxxxx | 1 | Xxxxxxxxx//xxxxxxxx//xxxxxx | | | | | | | | |
| J.O A TO INC | ALL ALL | 2 | Xxxxxxxxx//xxxxxxx//xxxxxx | | | | | | | | |
| | | 3 | Xxxxxxxxx//xxxxxxx//xxxxxx | | | | | | | | |
| | | 4 | Xxxxxxxxx//xxxxxxx//xxxxxx | | | | | | | | |
| | | 5 | Xxxxxxxxx//xxxxxxx//xxxxxx | | | | | | | | |
| | | 6 | Xxxxxxxxx//xxxxxxx//xxxxxx | | | | | | | | |

 $6.0 \times 10^6 \text{ hRPC}$ 

path\l\_program.sas date time

Programmer Note: sort by subject and AE # subject Programmer Note: include Onset Time if available in Onset Date column.

jCyte, Inc.
Protocol: JC-02

Listing 16.2.7.4
Post Injection Clinical Vitreous Exam
Safety Population

| | | | | Study Day | Not Done: Reason | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | | | Examination | | | Method | Cells | Change from | <u>l</u> | | | Photograph Taken? |
| Group | Subject ID | Visit | Date | | | Used | Visualized? | Prev. Visit | Appearance | Size | Location | |
| | | _ | | | | | | | | | | |
| Sham | XXXXXX | Day 0 | ISO8601 | XX | | Indirect | Yes/No | Yes/No | Cells | XXXXXX | XXXXXX | Yes/No |
| | | | | | | Ophthalmoscopy | | | | | | |
| | | Day 1 | | XX | | Fundus Exam | Yes/No | Yes/No | Clumps | XXXXXX | XXXXXX | Yes/No |
| | | Day 7 | | XX | | Slit Lamp Exam | Yes/No | Yes/No | Opacity | XXXXXX | XXXXXX | Yes/No |
| | | Day 28 | | | | Other: | Yes/No | Yes/No | Debris | XXXXXX | XXXXXX | Yes/No |
| | | Month 3 | | | | Fundus Exam | Yes/No | Yes/No | Inflammation | XXXXXX | XXXXXX | Yes/No |
| | | Month 6 | | | | | | | | | | |
| | | Month 9 | | | | Other: | Yes/No | Yes/No | Clumps | XXXXXX | XXXXXX | Yes/No |
| | | Month | | | | Indirect | Yes/No | Yes/No | Opacity | XXXXXX | XXXXXX | Yes/No |
| | | 12/Early | | | | Ophthalmoscopy | | | | | | |
| | | Termination | | | | | | | | | | |
| $3.0 \times 10^6$ hRPC | xxxxxx | Day 0 | | | | Indirect<br>Ophthalmoscopy | Yes/No | Yes/No | Cells | xxxxxx | xxxxxx | Yes/No |
| | | Day 1 | | | | Fundus Exam | Yes/No | Yes/No | Clumps | XXXXXX | XXXXXX | Yes/No |
| | | Day 7 | | | | Slit Lamp Exam | Yes/No | Yes/No | Opacity | XXXXXX | XXXXXX | Yes/No |
| | | Day 28 | | | | Other: | Yes/No | Yes/No | Debris | XXXXXX | XXXXXX | Yes/No |
| | | Month 3 | | | | Fundus Exam | Yes/No | Yes/No | Inflammation | XXXXXX | XXXXXX | Yes/No |
| | | Month 6 | | | | 1 011000 2110111 | 1 55/110 | 1 00,110 | | | | 1 00/110 |
| | | Month 9 | | | | Other: | Yes/No | Yes/No | Clumps | XXXXXX | XXXXXX | Yes/No |
| | | Month | | | | Indirect | Yes/No | Yes/No | Opacity | XXXXXX | XXXXXX | Yes/No |
| | | 12/Early | | | | Ophthalmoscopy | | | - [ | | | |
| | | Termination | | | | ориманновору | | | | | | |
| $6.0 \times 10^6$ | | 2 2111111111111111111111111111111111111 | | | | | | | | | | |
| hRPC | | | | | | | | | | | | |
| mu c | | | | | | | | | | | | |

path\l\_program.sas date time


Listing 16.2.8.1 Hematology Safety PopulationPart 1 of 2

| Treatmen<br>t Group | Subjec<br>ID | t<br>Visit | Collection<br>Date and<br>Time | Study Day | Not Done:<br>Reason | Lab Name | Hemoglobin<br>(g/dL) | Hematocrit | Platelet Count (x 10^9/L) | Red Cell Count<br>(x 10^12/L) | White Cell<br>Count<br>(x 10^9/L) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Sham | XXX | Screening | ISO8601 | XX | | UCI | | | | | |
| | | Baseline | ISO8601 | XX | | | | | | | |
| | | Day 28 | | XX | | | | | | | |
| | | Month 3 | | XX | | | | | | | |
| | | Month 6 | | XX | | | | | | | |
| | | Month | | XX | | | | | | | |
| | | 12/Early | | | | | | | | | |
| | | Terminatio | | | | | | | | | |
| | | n | | | | | | | | | |
| 3.0 x 10 <sup>6</sup><br>hRPC | XXX | Screening | | XX | | Lab Corp | | | | | |
| | | Baseline | | XX | | | | | | | |
| | | Day 28 | | XX | | | | | | | |
| | | Month 3 | | XX | | | | | | | |
| | | Month 6 | | XX | | | | | | | |
| | | Month | | XX | | | | | | | |
| | | 12/Early | | | | | | | | | |
| | | Terminatio | | | | | | | | | |
| | | n | | | | | | | | | |
| 6.0 x 10 <sup>6</sup><br>hRPC | xxx<br>xxx | | | | | | | | | | |

### Listing 16.2.8.1 Hematology Safety Population Part 2 of 2

Collection Study Not Done: Lab Neutro Lymph

| Treatment | Subject | | Date and | Day | Reason | Nam | phils | ocytes | Monocytes | Eosinophils | Basophils | Neutrophils | Lymphocytes | Monocytes | Eosinophils | Basophils |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | ID | Visit | Time | | | e | (%) | (%) | (%) | (%) | (%) | $(x 10^{9}/L)$ | $(x 10^9/L)$ | $(x 10^9/L)$ | $(x 10^9/L)$ | $(x 10^9/L)$ |

Sham UCI

Note: L=Low and H=High, CS=Clinically Significant

. path\l\_program.sas date time

Listing 16.2.8.2 Chemistry Safety Population Part 1 of 2

| | | | Collection | | Not | | | | | | Carbon | | | Alkaline | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatmen | Subject | | Date and | Study Day | Done: | Lab | Bilirubin | Sodium | Potassium | Chloride | Dioxide | ALT | AST | Phosphatase | HbA1c |
| t Group | ID | Visit | Time | | Reason | Name | (mg/dL) | (mmol/L)) | (mmol/L) | (mmol/L) | (mmol/L) | (U/L) | (U/L) | (U/L) | (%) |
| Sham | xxxxxx | Screening | ISO8601 | XX | | UCI | | | | | | | | | |
| | | Baseline | | XX | | | | | | | | | | | |

| Sham | XXXXXX | Screening | ISO8601 | XX | UCI |
|------|--------|-------------|---------|----|-----|
| | | Baseline | | XX | |
| | | Day 28 | | XX | |
| | | Month 3 | | XX | |
| | | Month 6 | | XX | |
| | | Month | | XX | |
| | | 12/Early | | | |
| | | Termination | | | |

 $3.0 \times 10^6 \times \text{xxx--xxx}$  Lab Corp hRPC

6.0 x 10<sup>6</sup> xxx--xxx hRPC

### Listing 16.2.8.2 Chemistry Safety PopulationPart 2 of 2

| Treatment<br>Group | Subject<br>ID | Visit | Collection Date and Time | Study Day | Not Done:<br>Reason | Lab Name | BUN<br>(mg/dL) | Creatinine (mg/dL) | Total Protein<br>(g/dL) | Albumin<br>(g/dL) | Calcium<br>(mg/dL) | Phosphate (mg/dL) | Glucose<br>(mg/dL) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sham | xxxxxx | Screening | ISO8601 | XX. | | UCI | | | | | | | |

Note: L=Low and H=High, CS=Clinically Significant.

path\l\_program.sas date time

### Listing 16.2.8.3 Urinalysis/Microscopic Exam Safety Population Part 1 of 2

| Treatment Group | Subject<br>ID | Visit | Collection<br>Date and<br>Time | Study Day | Not Done:<br>Reason | Lab Name | Specific<br>Gravity | рН | Glucose | Bilirubin | Ketone | Blood | Protein | Urobilinogen |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sham | XXX<br>XXX | Screening | ISO8601 | xx | | UCI | | | Negative | Negative | Negative | Negative | Negative | Negative |
| | | Baseline<br>Month 3<br>Month 6<br>Month12/Early<br>Termination | | | | | | | Negative<br>Negative<br>positive | Negative<br>Negative<br>positive | Negative<br>Negative<br>positive | Negative<br>Negative<br>positive | Negative<br>Negative<br>positive | Negative<br>Negative<br>positive |
| $3.0 \times 10^6 \text{ hRPC}$ | xxx-<br>xxx | | | | | Lab corp | | | | | | | | |
| $6.0 \times 10^6 \text{hRPC}$ | XXX | | | | | | | | | | | | | |

# Listing 16.2.8.3 Urinalysis/Microscopic Exam Safety Population Part 2 of 2

| N /I 1 | crosco | 110 | Hvom |
|--------|--------|-----|---------|
| IVII | CIUSCO | m | T/XaIII |

| | | | | | | | | N | Aicroscopic I | Exam | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Collection | | Not Done: | Lab Name | | | | | |
| Treatment | Subject | | Date and | | Reason | | WBC | RBC | <b>Epithelial</b> | | |
| Group | ΙĎ | Visit | Time | Study Day | | | (/hpf) | (/hpf) | Cells | Bacteria | Other |
| Sham | XXXXXX | Baseline | ISO8601) | XX | | UCI | | | Absent/Prese | Absent/Prese | |
| | | | | | | | | | nt | nt | |
| path\l_progra | am.sas date | time | | | | | | | | | |

### Listing 16.2.8.4 Clinically Significant Lab Values Safety Population

Collection

| Treatment Group | Subject ID | Visit | Collection Date and Time | Study Day | Lab Category | Lab Test | Value |
|---|---|---|---|---|---|---|---|
| Sham | xxxxxx<br> | Screening Baseline Day 28 Month 3 Month 6 Month 12/Early Termination | ISO8601<br>ISO8601 | xx<br>xx | Hematology | Hemoglobin<br>Hematocrit | |
| $3.0 \times 10^6 \text{hRPC}$ | xxxxxx | | | | | | |
| 6.0 x 10 <sup>6</sup> hRPC | xxxxxx | | | | Chemistry | Albumin | |

path\l\_program.sas date time

Programmer Note: Include only Clinically Significant Abnormal values from all Lab tests.

Listing 16.2.8.5 Coagulation Safety Population

Not Done: Reason Sample Analyzed Study Day Collection PT (sec) PTT (sec) INR at Local Treatment Group Subject ID Visit Laboratory Lab Name Date Sham ISO8601 Yes/No UCI Screening xxx--xxxXXxx xxx xXX XX  $3.0 \times 10^6 \, hRPC$ Yes/No UCI xxx--xxx Screening  $\mathbf{X}\mathbf{X}$ XX X XX X XX XX Screening  $6.0 \times 10^6 \, hRPC$ Yes/No UCI xx x xxx--xxx XXXX X XX XX

path\l program.sas date time

### Listing 16.2.8.6 Infectious Disease Assessments Safety Population

| Treatment Group | Subject ID | Visit | Collection Date and Time | Study Day | Not Done: Reason | Hepatitis B | Hepatitis C | HIV LAB Test |
|---|---|---|---|---|---|---|---|---|
| Sham | xxxxxx | Screening<br>Baseline | ISO8601<br>ISO8601 | XX | | Negative<br>Positive | Negative<br>Positive | Negative<br>Positive |
| $3.0 \times 10^6 \text{ hRPC}$ | XXXXXX | Screening<br>Baseline | ISO8601 | | | Not Done<br>Negative | Not Done<br>Negative | Not Done<br>Negative |
| $6.0 \times 10^6 \text{hRPC}$ | xxxxxx | Screening<br>Baseline | | | | Negative<br>Positive | Negative<br>Positive | Negative<br>Positive |

jCyte, Inc.
Protocol: JC-02

### Listing 16.2.8.7 HLA Typing Safety Population

| Treatment Group | Subject ID | HLA Typing Previously<br>Performed | If No, HLA Typing<br>Performed | Collection<br>Date | Study Day |
|---|---|---|---|---|---|
| Sham | XXXXXX | Yes/No | Yes/No | ISO8601 | XX |
| 3.0 x 10 <sup>6</sup> hRPC | xxxxxx | | | | |
| 6.0 x 10 <sup>6</sup> hRPC | xxxxxx | | | | |

path\l\_program.sas date

time

jCyte, Inc. Protocol: JC-02 Page 1 of x

Listing 16.2.8.8 Vital Signs Safety Population

| Treatment Group | Subject<br>ID | Visit | Measurement<br>Date and<br>Time | Study Day | Not Done: Reason | Time Point | SBP/DBP<br>(mmHg) | Heart Rate (beats/min) | Respiration<br>Rate<br>(breaths/min) | Temperature (°C) | Weight<br>(Kg) | Height<br>(cm) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sham | vvvvv | Screening | ISO8601 | XX | | | Xxx/xxx | XXX | XXX | xxx | XXX | xxx |
| Shum | AAA AAA | Baseline | 1500001 | XX | | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 | | XX | | 15 min Pre-Injection | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Duj 0 | | XX | | 15 min Post-Injection | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | | | XX | | 60 min Post-Injection | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 1 | | XX | | ov mm reev mjestien | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 7 | | XX | | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 28 | | XX | | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Month 3 | | XX | | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Month 6 | | XX | | | Xxx/xxx | xxx | XXX | XXX | XXX | XXX |
| | | Month 9 | | XX | | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | Month | | | | | | | | | | |
| | | 12/Early | | | | | | | | | | |
| | | Terminatio | ) | | | | | | | | | |
| | | n | | | | | | | | | | |
| 3.0 x 10 <sup>6</sup> hRPC | | Baseline | | XX | | | | | | | | |
| $6.0 \times 10^6 \text{ hRPC}$ | xxxxxx | Baseline | | XX | | | | | | | | |
| | | | | XX | | | Xxx/xxx | xxx | XXX | XXX | XXX | XXX |
| | | | | XX | | | Xxx/xxx | xxx | XXX | XXX | XXX | XXX |
| | | | | XX | | | Xxx/xxx | XXX | XXX | XXX | XXX | XXX |
| | | | | XX | | | Xxx/xxx | XXX | XXX | xxx | XXX | XXX |
| path\l_progra | m.sas date | time | | | | | | | | | | |

jCyte, Inc
Protocol No. JC-02

### Listing 16.2.8.9 Physical Examination Safety Population

| | | | | Study Day | Not Done: Reason | | ny Changes in Vision or Light<br>Perception since Prior Physical |
|---|---|---|---|---|---|---|---|
| Treatment | Subject | Visit | Examination | | | on the Physical | Examination |
| Group | IĎ | | Date | | | Exam? | |
| Sham | xxxxxx | Screening | ISO8601. | XX | | Yes/No | |
| | | Baseline | | XX | | Yes/No | |
| | | Day1 | ISO8601 | XX | | Yes/No | No |
| | | Day 7 | ISO8601 | XX | | Yes/No | Yes: Changes |
| | | Day 28 | ISO8601 | XX | | Yes/No | Yes: Changes |
| | | Month 3 | | | | | _ |
| | | Month 6 | | | | | |
| | | Month 12/Early | | | | | |
| | | Termination | | | | | |
| $3.0 \times 10^6 \text{ hRPC}$ | XXXXXX | | | | | | |
| 6.0 x 10 <sup>6</sup> hRPC | xxxxxx | | | | | | |

path\l\_program.sas date time

MPage 1 of x jCyte, Inc. Protocol: JC-02

### Listing 16.2.8.10 Prior and Concomitant Medications **Safety Population**

| Treatment Group | Subject<br>ID | CM<br># | Verbatim Term //<br>Preferred Drug Name//ATC Text 4 | Start Date and<br>Time<br>(Study Day) | Stop Date<br>(Study Day) | Dose | Units | Dose Form | Route | Frequency | Indication |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Sham | xxxxxx | 1 | Xxxxxxxxxxxx // xxxxxxxxxxx // xxxxxxxxx | ISO8601(xx) | ISO8601(xx) | xxx | mg | Tablet | Oral | Daily | MH#, AE#, injection procedure |
| | | 2 | Xxxxxxxxxxx // xxxxxxxxxx // | ISO8601(xx) | Ongoing | XXX | ug | Capsule | Oral | As Needed | procedure |
| | | 3 | Xxxxxxxxxxx // xxxxxxxxxx // xxxxxxxxxx | ISO8601(xx) | ISO8601(xx) | XX | ml | Suspension | Oral | Daily | |
| | | 4 | Xxxxxxxxxxxx // xxxxxxxxxxx // xxxxxxxxx | ISO8601(xx) | Ongoing | xxx | g | Ointment | Oral | Daily | |
| | | 5 | Xxxxxxxxxxxx // xxxxxxxxxxx // xxxxxxxxx | ISO8601(xx) | Ongoing | XX | Tablets | Tablet | Oral | Daily | |
| | | 6 | Xxxxxxxxxxxx // xxxxxxxxxxx // xxxxxxxxx | ISO8601(xx) | ISO8601(xx) | XXX | Capsules | Capsule | Oral | Daily | |
| | | 7 | Xxxxxxxxxxxx // xxxxxxxxxxx // xxxxxxxxx | ISO8601(xx) | Ongoing | XXX | Puff | Aerosol | Oral | 2X a Day | |
| | | 8 | Xxxxxxxxxxxx // xxxxxxxxxxx // xxxxxxxxx | ISO8601(xx) | ISO8601(xx) | XXX | mg | Powder | Oral | Every Month | |

.  $3.0 \times 10^6 \, hRPC$ XXX--XXX

 $6.0 \times 10^6 \, hRPC$ xxx--xxx

path\l\_program.sas date time

Programmer Note: sort by CM # within each subject.

jCyte, Inc
Protocol No. JC-02

Listing 16.2.8.11 Pregnancy Test Safety Population

| Treatment<br>Group | Subject<br>ID | Visit | Urine<br>Pregnancy<br>Collection Date | Study Day | Not Done:<br>Reason | Result | If Positive, Was a<br>Serum Test<br>Performed? | If Serum Test Performed,<br>Result |
|---|---|---|---|---|---|---|---|---|
| Sham | xxxxxx | Screening<br>Baseline<br>Month 12/<br>Early<br>Termination | ISO8601<br>ISO8601<br>ISO8601 | XX<br>XX<br>XX | | Positive/Negative<br>Positive/Negative<br>Positive/Negative | Yes/No | Positive/Negative<br>Positive/Negative<br>Positive/Negative |

.....

3.0 x 10<sup>6</sup> hRPC xxx--xxx

6.0 x 10<sup>6</sup> hRPC xxx--xxx

path\l\_program.sas date time

### **Listing 16.2.8.12** PRA and DRA Antibody Test Results **Safety Population**

| | | | | Study Day | |
|---|---|---|---|---|---|
| | Subject | | Collection | | Sample Collected: |
| Treatment Group | ID | Visit | Date and Time | | Reason |
| | | | | | _ |
| Sham | XXXXXX | Baseline | ISO8601 | XX | Yes/No: Reason |
| | | Day 28<br>Month12/Early<br>Termination | ISO8601 | XX | Yes/No: Reason |

 $3.0 \times 10^6 \text{ hRPC}$ XXX--XXX

 $6.0 \times 10^6 \text{ hRPC}$ XXX--XXX

path\l\_program.sas date time Protocol No. JC-02

# Listing 16.2.8.13.1 Slit Lamp Exam (OD) Safety Population Part 1 of 2

| Treatment<br>Group | Subject<br>ID | Visit | Exam<br>Date | Study Day | Not Done:<br>Reason | Eyelids | Change<br>from<br>Previous<br>Visit? | Eyelashes | Change<br>from<br>Previous<br>Visit? | Conjunctiva | Change from<br>Previous<br>Visit? | Sclera | Change<br>from<br>Previous<br>Visit? | Cornea | Change<br>from<br>Previous<br>Visit? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sham | XXXXX | x Screening<br>Baseline | IS08601<br>IS08601 | xx<br>xx | | Normal<br>Abnormal<br>CS | Yes:<br>Abnormal | Normal<br>Abnormal CS | Yes :<br>Abnormalit | Normal<br>Abnormal CS | Yes:<br>Abnormality | Normal<br>Abnormal<br>CS | Yes:<br>Abnormalit | Normal<br>Abnormal<br>t CS | Yes:<br>Abnormalit |
| | | Day 1 | IS08601 | XX | | Abnormal<br>NCS | ty<br>No | Abnormal NCS | y<br>S No | Abnormal NCS | S No | Abnormal<br>NCS | y<br>No | Abnormal<br>NCS | y<br>No |
| | | Day 7 | IS08601 | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Day 28 | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Month 3 | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| • | | Month 6 | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Month 9 | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Month | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | 12/Early | _ | | | | | | | | | | | | |
| | | Termination | ) | | | | | | | | | | | | |
| | | n | | | | | | | | | | | | | |
| 3.0 x 10 <sup>6</sup><br>hRPC | xxxxx | x Screening | | | | | | | | | | | | | |
| | | Baseline | | | | | | | | | | | | | |
| | | | | XX | | Abnormal<br>NCS | No | Abnormal NCS | S No | Abnormal NCS | S No | Abnormal<br>NCS | No | Abnormal<br>NCS | No |
| | | | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Month12/ | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | Early | | | | | | | | | | | | | |
| | | Termination | ) | | | | | | | | | | | | |
| | | n | | | | | | | | | | | | | |
| 3.0 x 10 <sup>6</sup><br>hRPC | XXXXX | x Screening | | | | | | | | | | | | | |
| ma c | | Baseline | | | | | | | | | | | | | |
| Note: CS | S=Clinica | ally Signific | ant, NCS=N | Not Clinically | Significant.pa | th\l_program. | sas date | e time | | | | | | | |


jCyte, Inc
Protocol No. JC-02

Part 2 of 2

Listing 16.2.8.13.1 Slit Lamp Exam (OD) Safety Population

| Treatment<br>Group | Subject<br>ID | | Exam<br>Date | Study Day | Not Done<br>:Reason | Anterior<br>Chamber<br>Flare | Change<br>from<br>Previous<br>Visit? | Iris | Change<br>from<br>Previous<br>Visit? | Lens Status | Cataract<br>Type | Catarac<br>Grade | Clinically<br>Significan<br>Findings<br>t for Grade | t | Other<br>Finding<br>Abnormalit | Change<br>from<br>ti Previou<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sham | xxx | Screening | ISO8601 | XX | | 0 | | Normal | | Aphakic | Nuclear | +1 | Yes/No | Finding: | Abnormal<br>CS | |
| | | Baseline | ISO8601 | XX | | +1 | Yes :<br>Abnorma<br>lity | Abnormal<br>CS | Yes :<br>Abnorma<br>lity | Psedophakic | Cortical | +2 | Yes/No | | | |
| | | Day 1 | ISO8601 | XX | | +1 | No | Abnormal<br>NCS | | Phakic | Posterior | +3 | Yes/No | | | |
| | | Day 7 | ISO8601 | XX | | +3 | | Normal | | Psedophakic | Nuclear | +1 | Yes/No | | | |
| | | Day 28 | ISO8601 | XX | | +4 | | Normal | | Phakic | Cortical | | Yes/No | | | |
| | | Month 3 | | XX | | +4 | | Normal | | Psedophakic | Nuclear | +4 | Yes/No | | | |
| | | Month 6 | | XX | | +1 | | Normal | | Phakic | Cortical | +1 | Yes/No | | | |
| | | Month 9 | | XX | | +4 | | Normal | | Aphakic | Posterior | +2 | Yes/No | | | |
| | | Month<br>12/Early | | XX | | +1 | | Normal | | Psedophakic | Nuclear | +3 | Yes/No | | | |
| | | Termination | ) | | | | | | | | | | | | | |
| | | n | | | | | | | | | | | | | | |
| 3.0 x 10 <sup>6</sup> → nRPC | xxxxxx | Screening | | | | | | | | | | | | | | |
| | | Baseline | | | | | | | | | | | | | | |
| | | | | XX | | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnorn<br>al NCS | | Abnormal<br>NCS | No | |
| | | | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | | |
| | | | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | | |
| | | | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | | |

Programmer Note: Listing 16.2.8.10.2 will contain the same information for the other eye (OS).
Protocol No. JC-02

### Listing 16.2.8.13.2 Slit Lamp Exam (OS) Safety Population Part 1 of 2

| Treatn<br>Grou | nent Su<br>up | | Visit | Exam<br>Date | Study<br>Day | Not Done:<br>Reason | Eyelids | Change<br>from<br>Previous<br>Visit? | Eyelashes | Change from<br>Previous<br>Visit? | Conjunctiva | Change from<br>Previous<br>Visit? | Sclera | Change from<br>Previous<br>Visit? | Cornea | Change from Previous Visit? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sham | | | Screening | gIS08601 | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | , | XXX | Baseline | IS08601 | XX | | Abnormal<br>CS | Yes :<br>Abnormal<br>ty | Abnormal<br>i CS | Yes:<br>Abnormality | Abnormal CS | Yes :<br>Abnormality | Abnormal CS | Yes :<br>Abnormality | | Yes : Abnormality |
| | | | Day 1 | IS08601 | XX | | Abnormal<br>NCS | | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No | Abnormal<br>NCS | No |
| | | | Day 7 | IS08601 | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | | Day 28 | IS08601 | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | | Month 3 | | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | | Month 6 | IS08601 | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | | Month 9 | IS08601 | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| | | | Month<br>12/Early<br>Terminat<br>on | IS08601<br>i | XX | | Normal | | Normal | | Normal | | Normal | | Normal | |
| 3.0 x 1<br>hRPC | | XX | Screening | gIS08601 | XX | | Normal | | Normal | | Normal | | Normal | | Normal | Baseline |
| mu c | • | | Baseline | IS08601 | XX | | Normal | | Normal | | Normal | | Normal | | Normal | Screening |

Note: CS=Clinically Significant, NCS=Not Clinically Significant..

path\l program.sas date

Programmer Note: Listing 16.2.8.10.2 will contain the same information for the other eye (OS).

Protocol No. JC-02

#### Listing 16.2.8.13.2 Slit Lamp Exam (OS) Safety Population Part 2 of 2

| Treatment Group | Subject<br>ID | Visit | Exam<br>Date | (Study<br>Day) | Not<br>Done:<br>Reason | Anterior<br>Chamber<br>Flare | Change<br>from<br>Previous<br>Visit? | Iris | Change from<br>Previous Visit? | Lens Status | Cataract<br>Type | Cataract<br>Grade | Clinically<br>Significant<br>Findings for<br>Grade ? | Other<br>Findings | Other<br>Finding<br>Abnormal<br>ties | Change<br>from<br>i Previous<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Sham | xxxxxx | Screening | ISO8601 | xx | | 0 | | Normal | | Aphakic | Nuclear | +1 | Yes/No | Finding: | Abnormal<br>CS | |
| | | Baseline | ISO860 | XX | | +1 | Yes :<br>Abnormal<br>ty | Abnormal CS<br>i | Yes:<br>Abnormality | Psedophaki<br>c | Cortical | +2 | Yes/No | | | |
| | | Day 1 | ISO860 | xx | | +1 | No | Abnormal<br>NCS | No | Phakic | Posterior | +3 | Yes/No | | | |
| | | Day 7 | ISO860 | XX | | +3 | | Normal | | Psedophaki<br>c | Nuclear | +1 | Yes/No | | | |
| | | Day 28 | ISO860 | XX | | +4 | | Normal | | Phakic | Cortical | +2 | Yes/No | | | |
| | | Month 3 | ISO860 | XX | | +4 | | Normal | | Psedophaki<br>c | Nuclear | +4 | Yes/No | | | |
| | | Month 6 | ISO860 | XX | | +1 | | Normal | | Phakic | Cortical | +1 | Yes/No | | | |
| | | Month 9 | ISO860 | XX | | +4 | | Normal | | Aphakic | Posterior | +2 | Yes/No | | | |
| | | Month<br>12/Early<br>Termination | ISO860 | XX | | +1 | | Normal | | Psedophaki<br>c | | +3 | Yes/No | | | |

 $3.0 \times 10^6$ XXX--XXX hRPC

 $6.0 \times 10^6$ XXX--XXX

hRPC

Note: CS=Clinically Significant, NCS=Not Clinically Significant.

path\l\_program.sas date time

Listing 16.2.8.14 Intraocular Pressure (IOP) Safety Population

| Treatment<br>Group | Subject<br>ID | Visit | Measurement Date and Time | Study Day | Not Done:<br>Reason | Device Used | OD (Right)<br>Mean IOP (mmHg) | OS (Left)<br>Mean IOP (mmHg) |
|---|---|---|---|---|---|---|---|---|
| Sham | xxxxxx | Baseline<br>Day 0 | ISO 8601<br>ISO 8601 | XX | | Tonopen | xx | XX |
| | | Day 0 | ISO 8601 | XX | | Tonopen | XX | XX |
| | | Day 7 | ISO 8601 | XX | | Other Device | XX | XX |
| | | Day 28 | ISO 8601 | XX | | | XX | XX |
| | | Month 3 | ISO 8601 | XX | | | XX | XX |
| | | Month 6 | ISO 8601 | XX | | | XX | XX |
| | | Month 9 | ISO 8601 | XX | | | XX | XX |
| | | Month | ISO 8601 | XX | | | XX | XX |
| | | 12/Early<br>Termination | | | | | | |
| 3.0 x 10 <sup>6</sup><br>hRPC | xxxxxx | Baseline | | | | | | |
| | | Day 0 Day 1 Day 7 Day 28 Month 3 Month 6 Month 9 Month 12/Early Termination | | | | | | |
| 6.0 x 10 <sup>6</sup><br>hRPC | xxxxxx | Baseline | | | | | | |

path\l\_program.sas date time

#### Listing 16.2.8.15 B-Scan Safety Population

| | | | | | | Stud | ly Eye | | Righ | t Eye (OD) | | | Left E | ye (OS) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatm | ı | | | | Not Done:<br>Reason | Injected<br>Cells<br>Visualized?i | | | Abnormal,<br>Change from<br>Previous | | Overall<br>Pathology Result | | Abnormal,<br>Change from<br>Previous | n Patholog<br>y | Overall<br>Pathology |
| ent | Subject | | Measurement | Study | | f Yes, | | B-Scan | Visit? | Observed | | B-Scan | Visit? | Result | Result |
| Group | ID | Visit | Date and Time | Day | | Description | Video Taken? | Result | | | | Result | | Observed | |
| Sham | xxxxxx | Baseline | ISO8601 | xx | | Yes:<br>Description/<br>No/NA | Yes/No/NA | Normal | Yes/No/NA | Retinal<br>Detachmen | Good/Poor<br>t | Normal | Yes/No/NA | Retinal<br>Detachm<br>ent | Good/Poor |
| | | Day 7<br>Month 6 | ISO8601<br>ISO8601 | XX | | Yes/No/NA | Yes/No/NA | Abnormal<br>CS:<br>Abnormali<br>ty | Yes/No/NA | Irregular<br>Posterior<br>detachment | Good/Poor | Abnormal<br>CS:<br>Abnormality | Yes/No/NA | Irregular<br>Posterior<br>detachme<br>nt | Good/Poor |
| | | Month 12/<br>Early<br>Termination | ISO8601 | XX | | Yes/No/NA | Yes/No/NA | | Yes/No/NA | | Good/Poor | Abnormal<br>NCS | Yes/No/NA | | Good/Poor |
| $3.0 \text{ x}$ $10^6$ hRPC | xxxxxx | Baseline | ISO8601 | XX | | Yes/No/NA | Yes/No/NA | Normal | Yes/No/NA | | Good/Poor | Normal | Yes/No/NA | | Good/Poor |
| | | Day 7<br>Month 6 | ISO8601<br>ISO8601 | xx | | Yes/No/NA | Yes/No/NA | Abnormal<br>CS:<br>Abnormali<br>ty | Yes/No/NA | | Good/Poor | Abnormal<br>CS:<br>Abnormality | Yes/No/NA | | Good/Poor |
| | | Month 12/<br>Early<br>Termination | ISO8601 | XX | | Yes/No/NA | Yes/No/NA | • | Yes/No/NA | | Good/Poor | Abnormal<br>NCS | Yes/No/NA | | Good/Poor |
| 6.0 x<br>10 <sup>6</sup><br>hRPC | | Baseline | | | | | | | | | | | | | |
| | CS=Clinica<br>program.s | | ant, NCS=Not Cl<br>time | inically S | ignificant. | | | | | | | | | | |
| Progra | mmer Not | e Include de | escription of abno | ormality c | and Clinically | Significant in | formation in " | B-Scan Resi | ılt" column. | | | | | | |


RUC Error! AutoText entry not defined.


RUC Error! AutoText entry not defined.

### Listing 16.2.8.16 Dilated Funduscopic Examination Safety Population Part 1 of 4

OD (Right) Not Done: Study Time of Examinati Day Reason If Abnormal, If Abnormal, Dilator Treatme on Change from Vitreous Change from Administrati Date and Subject Vitreous Previous Visit? Exam Optic Nerve Previous nt ID Visit Time Exam Results Severity Exam Visit? Optic Nerve Exam Severity Group on Sham xxx--xxx Screenin ISO8601 ISO8601 Normal Mild +1 Normal Mild+1 Baseline ISO8601 ISO8601 Not Done Moderate +2 Not Done Moderate +2 XX Day 1 ISO8601 ISO8601 Abnormal CS: Yes Severe +3 Abnormal Yes Severe +3 XX Abnormality CS: Abnormalit У Day 7 ISO8601 ISO8601 Abnormal NCS No Very Server Abnormal No Very Server +4 XX +4NCS Day 28 ISO8601 ISO8601 Normal Mild +1 Normal Mild +1 XX Month 3 ISO8601 ISO8601 XX Not Done Moderate +2 Not Done Moderate +2 Month 6 ISO8601 ISO8601 Abnormal CS: Yes Mild +1 Abnormal Yes Mild+1 XXAbnormality CS: Abnormalit У Month 9 ISO8601 XX Month Abnormal CS: Yes Abnormal Mild+1 ISO8601 XX Mild+1 Yes 12/Early CS: Abnormality Termina Abnormalit tion У ISO8601 Not Done Moderate+2 Not Done Moderate+2 3.0 xxxx--xxx Screenin XX  $10^{6}$ g hRPC Baseline ISO8601 Abnormal CS: Yes Mild+1 Abnormal Yes Mild+1 XX Abnormality CS: Abnormalit У Day 1 ISO8601 Abnormal NCS No Moderate+2 Abnormal No Moderate+2 XX NCS


Note: With respect to "Vitreous Exam", "Optic Nerve Exam", "Macula Exam", and "Peripheral Retina Exam" columns, CS=Clinically Significant, NCS=Not Clinically Significant.

path\l\_program.sas date time


Listing 16.2.8.16
Dilated Funduscopic Examination
Safety PopulationPart 2 of 4

OD (Right) Study Day Not Done: If Reason Abnormal, Time of Examinati Change If Abnormal, Dilator Macula from Peripheral Change from Peripheral on Macula Treatmen Subject Retina Exam Previous Visit? Retina Exam Administra Date and Exam Previous Exam t Group ID Visit tion Time Results Visit? Severity Results Severity Mild+1 Sham xxx--xxx Screening ISO8601 ISO8601 Normal Mild+1 Normal XXBaseline ISO8601 ISO8601 Not Done Moderate Not Done Moderate+2 XX+2Day 1 ISO8601 ISO8601 Abnormal Yes Severe+3 Abnormal CS: Yes Severe+3 XX CS: Abnormality Abnormalit y Very Server+4 Day 7 ISO8601 ISO8601 Abnormal No Very Abnormal No XX. . NCS Server+4 NCS Mild+1 Normal Mild+1 Day 28 ISO8601 ISO8601 XXNormal Month 3 ISO8601 ISO8601 Not Done Moderate Not Done Moderate+2 XX+2Month 6 ISO8601 ISO8601 Abnormal Yes Mild+1 Abnormal CS: Yes Mild+1 XXCS: Abnormality Abnormalit y Month 9 ISO8601 ISO8601 Not Done Mild+1 Month ISO8601 ISO8601 XX Not Done Mild+1 12/Early Terminatio n 3.0 x 10<sup>6</sup> xxx-xxx Screening ISO8601 ISO8601 Not Done Moderate Not Done Moderate+2 XXhRPC +2ISO8601 ISO8601 Severe+3 Abnormal CS: Mild+1 Baseline Abnormal Yes Yes XX CS: Abnormality Abnormalit ISO8601 Moderate Abnormal No Moderate+2 Day 1 Abnormal No XX NCS +2NCS Day 7



# Listing 16.2.8.16 Dilated Funduscopic Examination Safety Population Part 3 of 4

OS(Left)

| | | | | | | | | OS(1 | Leπ) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Time of | Examinat | Not | | | | | | |
| | | | Dilator | ion | Done | | If Abnormal, | | | If Abnormal, | Optic Nerv |
| Treatment | Subject | t | Adminis | Date and | Study Reas | son Exam | Change from | Vitreous Exam | Optic Nerve | Change from | Exam |
| Group | ID | Visit | tration | Time | Day | Results | Previous Visit? | Severity | Exam | Previous Visit? | Severity |
| Sham | XXX | Screening | n ISO860 | ISO8601 | XX | Normal | | Mild +1 | Normal | | Mild +1 |
| | AAA | | e ISO860 | ISO8601 | XX | Not Done | | Moderate +2 | Not Done | | Moderate + |
| | | Day 1 | _ | ISO8601 | XX | Abnormal<br>CS:<br>Abnormalit<br>y | Yes | Severe +3 | Abnormal<br>CS:<br>Abnormality | Yes | Severe +3 |
| | | Day 7 | 1 | ISO8601 | | Abnormal<br>NCS | No | Very Server +4 | NCS | No | Very Serve<br>+4 |
| | | Day 28 | ISO860 | ISO8601 | XX | Normal | | Mild +1 | Normal | | Mild +1 |
| | | Month 3 | 3 ISO860 | ISO8601 | XX | Not Done | | Moderate +2 | Not Done | | Moderate + |
| | | Month 6 | 6 ISO860<br>1 | ISO8601 | xx | Abnormal<br>CS:<br>Abnormalit<br>y | Yes | Mild +1 | Abnormal<br>CS:<br>Abnormality | Yes | Mild +1 |
| | | Month 9 | 9 ISO860<br>1 | ISO8601 | XX | Abnormal<br>NCS | No | Moderate +2 | Abnormal<br>NCS | No | Moderate + |
| | | Month<br>12/Early<br>Termina<br>tion | , | ISO8601 | XX | Not Done | | Mild +1 | Not Done | | Mild +1 |
| 3.0 x 10 <sup>6</sup> x<br>hRPC | xxx-xxx | x Screenii<br>g | n ISO860<br>1 | ISO8601 | XX | Abnormal<br>CS:<br>Abnormalit<br>y | Yes | Mild +1 | Abnormal<br>CS:<br>Abnormality | Yes | Mild +1 |
| | | Baseline | e ISO860<br>1 | ISO8601 | xx<br>xx | Abnormal<br>NCS | No | Not Done | Abnormal<br>NCS | No | Not Done |

| $6.0 \times 10^6$ | xxx-xxx Screenin ISO860 ISO8601 | XX | Not Done | | Moderate | Not Done | | Moderate |
|---|---|---|---|---|---|---|---|---|
| hRPC | g 1 | | | | | | | |
| | Baseline ISO860 ISO8601 | XX | Abnormal | Yes | Mild | Abnormal | Yes | Mild |
| | 1 | | CS: | | | CS: | | |
| | | | Abnormalit | | | Abnormality | | |
| | | | y | | | | | |
| | Time5. ISO8601 | XX | Abnormal | No | Moderate | Abnormal | No | Moderate |
| | | | NCS | | | NCS | | |

Note: With respect to "Vitreous Exam", "Optic Nerve Exam", "Macula Exam", and "Peripheral Retina Exam" columns, CS=Clinically Significant, NCS=Not Clinically Significant. path\\\_program.sas date time

Programmer Note: Sorting order is by  $W/2^{nd}$  injection,  $W/O2^{nd}$  injection, subject ID, examination date (include unscheduled visits in the date sequence), and examination time.

jCyte, Inc
Page 1 of x
Protocol No. JC-02

## Listing 16.2.8.16 Dilated Funduscopic Examination Safety Population Part 4 of 4

| | | | | <u>-</u> | | | | | | OS (Left) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatmen<br>t Group | Subject<br>ID | Visit | Time of<br>Dilator<br>Administrat<br>ion | Examination Date and Time | Study Day | Not Done:<br>Reason | Macula<br>Exam Results | If Abnormal,<br>Change from<br>Previous Visit? | Macula Exam<br>Severity | Peripheral Retina<br>Exam Results | If Abnormal,<br>Change from<br>Previous Visit? | Peripheral<br>Retina Exam<br>Severity |
| Sham | xxxxxx<br> | Screening<br>Baseline<br>Day 1 | ISO8601 | ISO8601<br>ISO8601<br>ISO8601 | xx<br>xx<br>xx | | Normal Abnormal CS: Abnormality | Yes | Mild +1<br>Moderate +2<br>Severe +3 | Normal<br>Not Done<br>Abnormal CS:<br>Abnormality | Yes | Mild +1<br>Moderate +2<br>Severe +3 |
| | | Day 7 | | ISO8601 | XX | | Abnormal NCS | No | Very Server+4 | Abnormal NCS | No | Very Server+4 |
| | | Day 28<br>Month 3<br>Month 6<br>Month 9<br>Month<br>12/Early<br>Terminati<br>on | | ISO8601<br>ISO8601<br>ISO8601<br>ISO8601<br>ISO8601 | xx<br>xx<br>xx<br>xx<br>xx | | Normal Abnormal CS: Abnormality Abnormal NCS | Yes<br>No | Mild+1<br>Moderate+2<br>Mild+1<br>Moderate+2<br>Mild+1 | Normal<br>Not Done<br>Abnormal CS:<br>Abnormality<br>Abnormal NCS<br>Not Done | Yes<br>No | Mild+1<br>Moderate+2<br>Mild+1<br>Moderate+2<br>Mild+1 |
| 3.0 x 10 <sup>6</sup><br>hRPC | xxxxxx | Screening | | ISO8601 | XX | | | | Moderate+2 | Not Done | | Moderate+2 |
| IIKPC | | Baseline | | ISO8601 | XX | | Abnormal CS: Abnormality | Yes | Mild+1 | Abnormal CS: Abnormality | Yes | Mild+1 |
| | | Day 1 | | ISO8601 | XX | | Abnormal NCS | No | Moderate+2 | Abnormal NCS | No | Moderate+2 |

Note: With respect to "Vitreous Exam", "Optic Nerve Exam", "Macula Exam", and "Peripheral Retina Exam" columns, CS=Clinically Significant, NCS=Not Clinically Significant.

path\\\_\text{program.sas} date \time

Programmer Note: Sorting order is by Sham,  $3.0 \times 10^6 \text{ hRPC}$ ,  $6.0 \times 10^6 \text{ hRPC}$ , subject ID, examination date (include unscheduled visits in the date sequence), and examination time.

jCyte, Inc
Protocol No. JC-02

Listing 16.2.8.17 Fundus Photographs Safety Population

| | | | _ | | Not Done: Reason |
|---|---|---|---|---|---|
| Treatment Group | Subject<br>ID | Visit | Date of Fundus Photographs Taken | Study Day | |
| Sham | xxxxxx | Baseline | ISO8601 | xx | |
| $3.0 \times 10^6 \mathrm{hRPC}$ | xxxxxx | Baseline | ISO8601 | xx | |
| 6.0 x 10 <sup>6</sup> hRPC | xxxxxx | Baseline | ISO8601 | xx | |

path\l\_program.sas date time


